CLINICAL TRIAL: NCT01572038
Title: A Multicenter, Open-Label, Single-Arm Study of Pertuzumab in Combination With Trastuzumab and a Taxane in First Line Treatment of Patients With HER2-Positive Advanced (Metastatic or Locally Recurrent) Breast Cancer
Brief Title: A Study of Pertuzumab in Combination With Trastuzumab (Herceptin) and a Taxane in First-Line Treatment in Participants With Human Epidermal Growth Factor 2 (HER2)-Positive Advanced Breast Cancer
Acronym: PERUSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO28047; 2011-005334-20 (EudraCT Number)
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; 130-nm albumin-bound paclitaxel; Paclitaxel; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pertuzumab + Trastuzumab + Taxane (Experimental): Participants will receive pertuzumab and trastuzumab (Herceptin) IV plus a taxane in cycles of 3 weeks each until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurs first. Taxane chemotherapy can be either docetaxel, paclitaxel or nab-paclitaxel as per investigator's choice.
  Interventions: Drug: Docetaxel; Drug: Nab-paclitaxel; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Docetaxel — Participants may receive 'docetaxel' taxane chemotherapy as per investigator's choice, administered in line with the respective product information and/or recognized clinical practice guidelines.
Drug: Nab-paclitaxel — Participants may receive 'nab-paclitaxel' taxane chemotherapy as per investigator's choice, administered in line with the respective product information and/or recognized clinical practice guidelines.
Drug: Paclitaxel — Participants may receive 'paclitaxel' taxane chemotherapy as per investigator's choice, administered in line with the respective product information and/or recognized clinical practice guidelines.
Drug: Pertuzumab — Participants will receive pertuzumab 840 milligrams (mg) IV on Day 1 or Day 2 of Cycle 1, followed by 420 mg IV on Day 1 or Day 2 of each subsequent 3-week cycle.
  Other Names: RO 43-68451
Drug: Trastuzumab — Participants will receive trastuzumab (Herceptin) 8 milligrams per kilogram (mg/kg) IV on Day 1 or Day 2 of Cycle 1, followed by 6 mg/kg IV on Day 1 or Day 2 of each subsequent 3-week cycle, administered in line with the respective product Information and/or recognized clinical practice guidelines.
  Other Names: Herceptin

SUMMARY:
This multicenter, open-label, single-arm, Phase IIIb study will evaluate the safety and tolerability of pertuzumab in combination with trastuzumab (Herceptin) and a taxane (docetaxel, paclitaxel or nab-paclitaxel) in first-line treatment in participants with metastatic or locally recurrent HER2-positive breast cancer. Participants will receive pertuzumab intravenously (IV) and trastuzumab (Herceptin) IV plus a taxane in cycles of 3 weeks each until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with metastatic or locally recurrent disease not amenable to curative resection
* HER2-positive breast cancer
* Eastern cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* LVEF of at least 50 percent (%)

Exclusion Criteria:

* Previous systemic non-hormonal anti-cancer therapy for metastatic or locally recurrent disease
* Disease-free interval from completion of adjuvant or neoadjuvant systemic non-hormonal treatment to recurrence less than or equal to (</=) 6 months
* Previous approved or investigative anti-HER2 agents in any breast cancer treatment setting, except for trastuzumab and/or lapatinib in the adjuvant or neoadjuvant setting
* Disease progression while receiving trastuzumab and/or lapatinib in the adjuvant or neoadjuvant setting
* History of persistent Grade 2 or higher (National Cancer Institute Common Toxicity Criteria [NCI-CTC], Version 4.0) hematological toxicity resulting from previous adjuvant or neoadjuvant therapy
* Central nervous system (CNS) metastases
* Current peripheral neuropathy of Grade 3 or greater (NCI-CTC, version 4.0)
* History of other malignancy within the last 5 years prior to first study drug administration, except for carcinoma in situ of the cervix or basal cell carcinoma
* Inadequate bone marrow, liver or renal function
* Uncontrolled hypertension
* Hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1436 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (299):
- CPMC; Service d'Oncologie Médicale, Algiers, Algeria
- Argentina (2):
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Instituto de Oncología de Rosario, Rosario
- Australia (6):
  - Canberra Hospital; Medical Oncology, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital; Medical Oncology, Camperdown, New South Wales
  - HOCA Chermside, Chermside, Queensland
  - Mater Hospital; Cancer Services, South Brisbane, Queensland
  - Austin and Repatriation Medical Centre; Cancer Services, Melbourne, Victoria
  - Royal Melbourne Hospital; Hematology and Medical Oncology, Parkville, Victoria
- Austria (8):
  - Lkh-Univ. Klinikum Graz; Klinik Für Gynäkologie, Graz
  - LKH-UNIV. KLINIKUM GRAZ; Klinische Abteilung für Onkologie, Graz
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Abt. Für Gynäkologie, Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern; Abt. fur Innere Medizin 1, Linz
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - A.Ö. Lhk; Ii. Medizinische Abt. Mit Schwerpunkt Gaströnter. & Onkologie, Steyr
  - Medizinische Universität Wien; Univ.Klinik für Frauenheilkunde - Klinik für Gynäkologie, Vienna
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Abt. für Onkologie, Vienna
- Belgium (5):
  - UZ Brussel, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
- Brazil (7):
  - Oncologistas Associados, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital Sirio Libanes; Centro de Oncologia, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
- Canada (10):
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Bcca - Vancouver Island Cancer Centre; Oncology, Victoria, British Columbia
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - William Osler Health System Brampton Civic Hospital, Brampton, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - CSSS champlain - Charles-Le Moyne, Greenfield Park, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- China (9):
  - Beijing Cancer Hospital, Beijing
  - Southwest Hospital , Third Military Medical University, Chongqing
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Heilongjiang Provincial Tumor Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - The First Affiliated Hospital of The Fourth Military Medical University (Xijing Hospital), Xi'an
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
- Ecuador (2):
  - Hospital Solca Portoviejo; Oncologia, Portoviejo
  - Hospital Solca Quito; Oncologia, Quito
- Egypt (3):
  - Manial Specialized Hospital; Oncology, Cairo
  - El Mokatam HIO Hospital, Cairo
  - Nci; Oncology Dept, Cairo
- Estonia (2):
  - North Estonia Medical Centre Foundation; Oncology Center, Tallinn
  - Tartu University Hospital; Clinic of Hematology and Oncology, Tartu
- Finland (4):
  - Helsinki University Central Hospital; Oncology Clinics, Helsinki
  - Satakunta Central Hospital; Oncology, Pori
  - Tampere University Hospital; Dept of Oncology, Tampere
  - Turku Uni Central Hospital; Oncology Clinics, Turku
- France (29):
  - Clinique De L Europe; Radiotherapie Chimiotherapie, Amiens
  - ICO Paul Papin; Oncologie Medicale., Angers
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Centre Hospitalier Fleyriat; Oncologie/Hematologie, Bourg-en-Bresse
  - Centre Leonard De Vinci;Chimiotherapie, Dechy
  - Fondation Clement Drevon; Oncology, Dijon
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Clinique Sainte Marguerite; Oncologie Medicale, Hyères
  - Polyclinique de Blois; Chimiotherapie Ambulatoire, La Chaussée-Saint-Victor
  - Clinique Victor Hugo, LeMans
  - Polyclinique Du Bois; Centre Bourgogne, Lille
  - Clinique Chenieux; Oncology, Limoges
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Paoli Calmettes; Oncologie Medicale, Marseille
  - Centre Azureen De Cancerologie; Cons externes, Mougins
  - Hopital Cochin; Unite Fonctionnelle D Oncologie, Paris
  - Hopital Hotel Dieu; Oncologie Medicale, Paris
  - Institut Curie; Oncologie Medicale, Paris
  - Hopital Saint Louis; Service Onco Thoracique, Paris
  - Centre Catalan D' Oncologie, Perpignan
  - Polyclinique De Courlancy; Centre Radiotherapie Oncologie, Reims
  - Centre Eugene Marquis; Unite Huguenin, Rennes
  - Centre Rene Huguenin; ONCOLOGIE GENETIQUE, Saint-Cloud
  - Chp Saint Gregoire; Cancerologie Radiotherapie, Saint-Grégoire
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Institut D Oncologie Medical, Strasbourg
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Hopital Prive Drome Ardeche; Hopital De Jour, Valence
  - Clinique Onco Des Dentellieres; Chimiotherapie Radiotherapie, Valenciennes
- Germany (20):
  - Klinikum am Bruderwald; Frauenklinik, Bamberg
  - Gynaekologicum Bremen; Prof. Dr. Willibald Schröder, Bremen
  - Universitätsklinikum Erlangen; Frauenklinik, Erlangen
  - Universitätsklinikum Essen; Zentrum Für Frauenheilkunde, Essen
  - Klinikum Esslingen; Klinik für Frauenheilkunde und Geburtshilfe, Esslingen am Neckar
  - AGAPLESION Markus-Krankenhaus, Frankfurt
  - SRH Wald-Klinikum Gera; Klinik für Frauenheilkunde und Geburtshilfe, Gera
  - Universitätsklinikum Hamburg-Eppendorf; Frauenklinik, Hamburg
  - Gynaekologisch-Onkologische Schwerpunktpraxis Prof. Dr. med. Lueck, Dr. Schrader und Dr. Noeding, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes; Klinik f. Frauenheilkunden und Geburtshilfe, Homburg/Saar
  - St.-Vincenz-Krankenhaus; Frauenklinik, Limburg
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Brustzentrum Rhein-Ruhr Servicegesellschaft mbH, Mönchengladbach
  - Klinikum rechts der Isar der TU München; Klinik und Poliklinik für Frauenheilkunde, München
  - Ruppiner Kliniken, Klinik fuer Gynaekologie und Geburtshilfe, Neuruppin
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme)
  - Praxis Dr. Wagner, Saarbrücken
  - Kreiskrankenhaus Torgau; Abt.Gynäkologie und Geburtshilfe, Torgau
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
- Greece (7):
  - Anticancer Hospital Ag. Savas ; 2Nd Dept. of Oncology - Internal Medicine, Athens
  - Hippokratio Hospital; 2Nd Internal Medicine, Athens
  - University General Hospital of Heraklion, Crete
  - University Hospital of Larissa; Oncology, Larissa
  - University Hospital of Patras Medical Oncology, Pátrai
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- Queen Elizabeth Hospital; Clinical Oncology, Hong Kong, Hong Kong
- Hungary (6):
  - Szent Margit Hospital; Dept. of Oncology, Budapest
  - Fovarosi Szent Laszlo Korhaz-Rendelointezet; Onkologiai Osztaly X, Budapest
  - Orszagos Onkologial Intezet; Onkologiai Osztaly X, Budapest
  - Debreceni Egyetem Klinikai Kozpont ; Department of Oncology, Debrecen
  - Borsod-Abauj-Zemplen Megyei Korhaz Es Egyetemi Oktato Korhaz; Onkologiai Osztaly, Miskolc
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
- Israel (12):
  - Soroka Medical Center; Oncology Dept, Beersheba
  - Rambam Medical Center; Oncology, Haifa
  - Wolfson Hospital; Oncology, Holon
  - Shaare Zedek Medical Center; Oncology Dept, Jerusalem
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Nahariya Hospital; Oncology, Nahariya
  - Rabin Medical Center; Oncology Dept, Petah Tikva
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
  - Kaplan Medical Center; Oncology Inst., Rehovot
  - Sourasky / Ichilov Hospital; Dept. of Oncology, Tel Aviv
  - Assuta Medical Centre; Oncology, Tel Aviv
  - Assaf Harofeh; Oncology, Ẕerifin
- Italy (19):
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino, Campania
  - Az. Osp. Ospedale Civile; U.O. Di Oncologia Medica Ed Ematologia, Piacenza, Emilia-Romagna
  - Azienda USL di Ravenna; Unità Operativa di Oncologia Medica, Ravenna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria Dipartimento Interaziendale Di Oncologia, Udine, Friuli Venezia Giulia
  - Ospedale Belcolle Di Viterbo; Oncologia, Viterbo, Lazio
  - Ente Ospedaliero Ospedali Galliera; S.C. Oncologia Medica, Genoa, Liguria
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - Ospedale Mater Salutis; Dept of Oncology, Legnago, Lombardy
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Irccs Policlinico S. Matteo - Uni Pavia; Clinica Medica I Div. Med. Int. Onc. Medica E Gastroent., Pavia, Lombardy
  - Ospedale Maggiore Della Carita; Oncologia Medica, Novara, Piedmont
  - Ospedale Degli Infermi Di Biella; Reparto Oncologia Medica, Ponderano (BI), Piedmont
  - Fondazione Del Piemonte; Medical Oncology, Turin, Piedmont
  - Ospedale S. Vincenzo; Oncologia Medica, Taormina, Sicily
  - Ospedali Riuniti Di Ancona; Oncology, Ancona, The Marches
  - Ospedale Di Macerata; Oncologia, Macerata, The Marches
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
  - Arcispedale S.Anna; Oncologia Medica, Cona (Ferrara), Veneto
- Lebanon (2):
  - American University of Beirut - Medical Center, Beirut
  - Hotel Dieu de France; Oncology, Beirut
- Lithuania (2):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Uni Oncology Inst. ; Chemo - Radiation Dept, Vilnius
- Mexico (8):
  - Iem-Fucam, D.F.
  - Medica Sur Centro Oncologico Integral, D.F.
  - Instituto Nacional de Cancerologia; Oncology, Distrito Federal
  - Consultorio de Medicina Especializada; Dentro de Condominio San Francisco, Mexico City
  - Centro Medico Nacional Siglo Xxi - Imss; Hospital de Oncologia, Mexico City
  - Hospital General de México; Unidad de Oncologia, Mexico City
  - Instituto Nacional de Ciencias Médicas Y de La Nutricion Zubirán, Mexico City
  - Cancerologia de Queretaro; Oncologia, Queretaro, Queretaro
- Institut National D'oncologie Sidi Mohammed Ben Abdellah; Anatomopathologie, Rabat, Morocco
- Netherlands (8):
  - Medisch Centrum Alkmaar, Alkmaar
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina ZKHS; Inwendige Geneeskunde Afd., Eindhoven
  - Martini Ziekenhuis; Dept of Internal Medicine, Groningen
  - Mc Haaglanden, Locatie Antoniushove; Interne Geneeskunde, Leidschendam
  - Ikazia Ziekenhuis; Interne Oncologie, Rotterdam
  - Twee Steden Ziekenhuis - Locatie Tilburg; Interne Geneesekunde, Tilburg
  - Vie Curie, Venlo
- Pakistan (3):
  - Shifa International Hospital; Department of Oncology, Islamabad
  - Shaukat Khanum Memorial Cancer Hospital; Department of Oncology, Lahore
  - Hameed Latif Hospital; Department of Oncology, Lahore
- Peru (3):
  - Instituto;Oncologico Miraflores, Lima
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
  - Hospital Nacional LNS dela Policia Nacional del Perú. Unidad Onco; Deapartamento de Oncología, Lima
- Poland (6):
  - Bialostockie Centrum Onkologii; Oddzial Onkologii Klinicznej, Bialystok
  - Świętokrzyskie Centrum Onkologii; Dział Chemioterapii, Kielce
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii; Poradnia Chemioterapii, Lodz
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Cent.Onkologii-Instytut im. M. S-Curie, Klinika Now. Piersi i Chirurgii Rekon, Warsaw
- Portugal (8):
  - IPO de Coimbra; Servico de Oncologia Medica, Coimbra
  - Hospital do Espirito Santo; Servico de Oncologia Medica, Evora
  - Centro Clinico Champalimaud; Oncologia Medica, Lisbon
  - Hospital da Luz; Departamento de Oncologia Medica, Lisbon
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - Hospital Beatriz Angelo; Departamento de Oncologia, Loures
  - IPO do Porto; Servico de Oncologia Medica, Porto
  - Hospital de Sao Joao; Servico de Oncologia, Porto
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Centre; Oncology, Riyadh
  - King Abdul Aziz Medical City, King Fahd National Guard; Oncology, Riyadh
- Serbia (2):
  - Institute for Onc/Rad Serbia, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Spain (48):
  - Hospital Virgen de los Lirios; Servicio de Oncologia, Alcoy, Alicante
  - Hospital General de Elda; Servicio de Oncologia, Elda, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital de Jerez de la Frontera; Servicio de Oncologia, Jerez de la Frontera, Cadiz
  - Hospital Provincial de Castellon; Servicio de Oncologia, Castellon, Castellon
  - Hospital de Barbastro; Servicio de Oncologia, Barbastro, Huesca
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Complejo Hospitalario San Millan - San Pedro; Servicio de Oncologia, Logroño, La Rioja
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital de Gran Canaria Dr. Negrin; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Fundacion Hospital de Alcorcon; Servicio de Oncologia, Alcorcón, Madrid
  - Hospital Severo Ochoa; Servicio de Oncologia, Leganés, Madrid
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital de Cabueñes; Servicio de Oncologia, Gijón, Principality of Asturias
  - Hospital Universitari Sant Joan de Reus; Servicio de Oncologia, Reus, Tarragona
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Oncologia, Santa Cruz de Tenerife, Tenerife
  - Hospital de Sagunto; Servicio de Oncologia, Sagunto, Valencia
  - Hospital de Basurto; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital Quiron Barcelona; Servicio de Oncologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Complejo Asistencial Universitario De Burgos; Servicio de Oncologia, Burgos
  - Hospital San Pedro De Alcantara; Servicio de Oncologia, Cáceres
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Oncologia, Girona
  - Hospital Universitario Virgen de las Nieves; Servicio de Oncologia, Granada
  - Hospital General Universitario de Guadalajara; Servicio de Oncologia, Guadalajara
  - Complejo Asistencial Universitario de Leon; Servicio de Oncologia, León
  - Centro Oncologico MD Anderson Internacional; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Fundacion Jimenez Diaz; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Oncologia, Murcia
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Complejo Hospitalario de Orense; Servicio de Oncologia, Ourense
  - Hospital Clinico Universitario de Salamanca; Servicio de Oncologia, Salamanca
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Clinico Universitario de Valladolid; Servicio de Oncologia, Valladolid
  - Hospital de Rio Hortega; Servicio de Oncologia, Valladolid
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Oncologia, Zaragoza
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (6):
  - Gävle Sjukhus; Onkologiska Kliniken, Gävle
  - Sahlgrenska Universitetssjukhuset; Jubileumskliniken, Gothenburg
  - Centralsjukhuset Karlstad, Onkologkliniken, Karlstad
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Centrallasarettet Växjö, Onkologkliniken, Vaxjo
  - Västmanlands sjukhus Västerås, Onkologkliniken, Västerås
- Turkey (Türkiye) (5):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital; Medical Oncology, Adana
  - Akdeniz University Medical Faculty; Medical Oncology Department, Antalya
  - Ege University Medical Faculty; Medical Oncology Department, Bornova, İ̇zmi̇r
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara
- Ukraine (4):
  - Mun. Multifield Clin.Hosp.#4,Dept. of Chemotherapy, DSMU; Chair of Oncology and Medical Radiology, Dnipropetrovsk
  - Kyiv City Clinical Oncological Center; Chemotherapy Department, Kiev
  - State Oncology Regional Treatment-Diagnostic Center; Chemotherapy Department, Lviv
  - Zaporozhye Regional Oncology Hospital; Dept of Oncology, Zaporizhzhya
- Tawam Hospital, Al Ain City, United Arab Emirates
- United Kingdom (31):
  - Royal United Hospital; Oncology Department, Bath
  - City Hospital NHS Trust, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrookes Hospital; Dept of Oncology, Cambridge
  - Velindre Hospital, Cardiff
  - Walsgrave Hospital, Coventry
  - Royal Derby Hospital, Derby
  - University Hospital of North Durham, Durham
  - Hairmyres Hospital; Oncology Dept, East Kilbride
  - Eastbourne District Hospital; Department of Pharmacy, Eastbourne
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Diana Princess of Wales Hosp., Grimsby
  - Royal Surrey County Hospital, Guildford
  - Leeds Teaching Hosp NHS Trust;St James's Institute of Onc, Leeds
  - Huddersfield Royal Infirmary - Pharmacy department, Lindley
  - Barts and the London NHS Trust., London
  - Royal Free Hospital; Dept of Oncology, London
  - Kings College Hospital NHS Foundation Trust, London
  - Royal Marsden Hospital - London, London
  - Macclesfield District General Hospital, Macclesfield
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - James Cook Uni Hospital, Middlesbrough
  - Freeman Hospital; Northern Centre For Cancer Care, New Castle Upon Tyne
  - Mount Vernon Cancer Centre, Northwood
  - Churchill Hospital, Oxford
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital; Plymouth Oncology Centre, Plymouth
  - Musgrove Park Hospital, Somerset
  - The Royal Marsden Hospital, Sutton
  - Royal Cornwall Hospital, Truro
  - Wishaw General Hospital, Wishaw
- Uruguay (3):
  - Grupo Oncológico Cooperativo Uruguayo; Hospital de Clínicas - Dpto. de Oncología, Montevideo
  - Hospital Central De Las FF.AA.; Servicio De Oncologia, Montevideo
  - Hospital Pereira Rossell; Oncology Department, Montevideo
- Venezuela (2):
  - Centro Integral de Oncología, Caracas
  - Centro Médico Docente La Trinidad; Servicio de Gastroenterología, Caracas

REFERENCES:
- [Derived] Bachelot T, Ciruelos E, Schneeweiss A, Puglisi F, Peretz-Yablonski T, Bondarenko I, Paluch-Shimon S, Wardley A, Merot JL, du Toit Y, Easton V, Lindegger N, Miles D; PERUSE investigators. Preliminary safety and efficacy of first-line pertuzumab combined with trastuzumab and taxane therapy for HER2-positive locally recurrent or metastatic breast cancer (PERUSE). Ann Oncol. 2019 May 1;30(5):766-773. doi: 10.1093/annonc/mdz061. PMID 30796821

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1697 patients were screened: 261 failed screening and 1436 were enrolled in the study.
Groups:
- Pertuzumab + Trastuzumab + Taxane: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Taxane chemotherapy was docetaxel, paclitaxel, or nab-paclitaxel, per the investigator's choice.
Period: Overall Study
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Started (Intent-to-Treat (ITT) Population) | 1436 (All participants who were enrolled in the study.)
Received at Least One Dose of Study Drug (Safety Population) | 1436
Completed | 445
Not Completed | 991
Not completed — Death | 648
Not completed — Withdrawal by Subject | 204
Not completed — Lost to Follow-up | 81
Not completed — Physician Decision | 20
Not completed — Patient Decision | 14
Not completed — Progressive Disease | 8
Not completed — Site Closed Before Completing Form | 6
Not completed — Enrolled into Another Trial | 3
Not completed — Participated in Another Trial | 3
Not completed — Termination by Sponsor | 2
Not completed — Patient Deterioration | 1
Not completed — Sponsor Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1429
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1032
  Black | 9
  Asian | 88
  Native American | 28
  Other | 57
  Not Applicable as per Local Regulations | 222
Age Categorical (≤65 or >65 Years Old) [Count of Participants; unit: Participants]
  ≤65 Years Old | 1167
  >65 Years Old | 269
Ethnicity [Count of Participants; unit: Participants]
  Hispanic/Latino | 269
  Chinese | 57
  Japanese | 2
  Mixed Ethnicity | 18
  Indian | 21
  Other | 495
  Not Applicable as per Local Regulations | 574
Geographic Region of Enrollment [Count of Participants; unit: Participants] — Geographic region of enrollment was categorized as follows: Europe = Austria, Belgium, Estonia, Finland, France, Germany, Greece, Hungary, Italy, Lithuania, Netherlands, Poland, Portugal, Serbia, Slovenia, Spain, Sweden, United Kingdom, Ukraine; Asia = China, Hong Kong, Israel, Lebanon, Pakistan, Saudi Arabia, Turkey, United Arab Emirates; North America = Canada; South America = Argentina, Brazil, Ecuador, Mexico, Peru, Uruguay, Venezuela; Africa = Algeria, Egypt, Morocco; and Other = Australia.
  Participants
    Europe | 1009
    Asia | 177
    North America | 34
    South America | 121
    Africa | 71
    Other (Australia) | 24
Eastern Cooperative Oncology Group (ECOG) Performance Status at Baseline [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; Grade 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    Grade 0 or 1 | 1371
    Grade 2 | 63
    Missing | 2
Visceral Disease at Baseline [Count of Participants; unit: Participants] — The disease was considered as "visceral" if at least one lesion in a location other than breast, bone, bone marrow, lymph nodes, skin and soft tissue was observed during baseline tumor assessment. The disease was considered as "non-visceral" if all lesions observed at baseline were localized in breast, bone, bone marrow, lymph nodes, skin and soft tissue.
  Participants
    Visceral Disease | 992
    Non-visceral Disease | 444
Hormone Receptor Status of Disease at Baseline [Count of Participants; unit: Participants] — Hormone receptor status of the primary tumor and metastatic disease (combined) was defined as follows: Positive: if either estrogen receptor (ER) or progesterone receptor (PgR) status was positive; Negative: if both ER and PgR status was negative; Unknown: if both the ER and PgR status was unknown.
  Participants
    Positive | 918
    Negative | 512
    Unknown | 6
Prior Neoadjuvant or Adjuvant Chemotherapy Received [Count of Participants; unit: Participants]
  Prior (Neo)Adjuvant Chemotherapy | 786
  No Prior (Neo)Adjuvant Chemotherapy | 650
Previous Trastuzumab Therapy Received for Breast Cancer [Count of Participants; unit: Participants]
  Previous Trastuzumab Therapy | 400
  No Previous Trastuzumab Therapy | 1036
Initial Type of Taxane Received During the Study: Docetaxel, Paclitaxel, or Nab-Paclitaxel [Count of Participants; unit: Participants]
  Docetaxel | 775
  Paclitaxel | 588
  Nab-Paclitaxel | 65
  None | 8
Measurable or Non-Measurable Disease (per RECIST v1.1) at Baseline [Count of Participants; unit: Participants]
  Measurable Disease | 1198
  Non-Measurable Disease | 238

OUTCOME MEASURES:

1. Primary Outcome: Overview of the Number of Participants With at Least One Treatment-Emergent Adverse Event, Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0)
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. TEAEs to monitor included anaphylaxis and hypersensitivity, cardiac dysfunction, diarrhoea Grade ≥3, pregnancy-related AEs, interstitial lung disease, infusion-/administration-related reactions, mucositis, (febrile) neutropenia, rash/skin reactions, and suspected transmission of infectious agent. TEAEs of special interest included LVEF decreased, liver enzymes increased, and suspected transmission of infectious agent by the study drug.
Time Frame: From Baseline until 28 days after, or 7 months after (only for serious AEs related to study drug), the last dose of study treatment. The median (full range) duration of exposure to any study treatment was 16.2 (0.0-86.4) months.
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any TEAE - Any Grade | 1419
  Any TEAE - Grade 3 or Higher (≥3) | 879
  Any Serious TEAE | 535
  Any TEAE Leading to Death | 31
  Any TEAE Related to Pertuzumab - Any Grade | 1037
  Any TEAE Related to Trastuzumab - Any Grade | 946
  Any TEAE Related to Taxane - Any Grade | 1342
  Any TEAE Related to Pertuzumab - Grade ≥3 | 286
  Any TEAE Related to Trastuzumab - Grade ≥3 | 245
  Any TEAE Related to Taxane - Grade ≥3 | 514
  Any TEAE Leading to Interruption of Pertuzumab | 334
  Any TEAE Leading to Interruption of Trastuzumab | 386
  Any TEAE Leading to Interruption of Taxane | 354
  Any TEAE Leading to Discontinuation of Pertuzumab | 140
  Any TEAE Leading to Discontinuation of Trastuzumab | 133
  Any TEAE Leading to Discontinuation of Taxane | 286
  Any TEAE to Monitor - Any Grade | 1320
  Any TEAE to Monitor - Grade ≥3 | 535
  Any TEAE of Special Interest | 91
  Any TEAE Within 28 Days of Treatmt Discontinuation | 975

2. Primary Outcome: Number of Participants Who Died Over the Course of the Study by Reported Cause of Death (Adverse Events Leading to Death by System Organ Class and Preferred Term)
Description: All adverse events leading to death, regardless of whether they were classified as treatment emergent, are listed by system organ class (SOC) and preferred term (PT) according to the Medical Dictionary for Regulatory Activities, version 22.1 (MedDRA version 22.1); PTs that are part of a given SOC are listed in the rows directly below each SOC within the results table. Admin. = administration; Mediast. = mediastinal
Time Frame: The median (full range) duration of follow-up was 68.73 (0.03-87.29) months.
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Total Number of Deaths | 658
  Number of Deaths by Cause: Progressive Disease | 581
  Number of Deaths by Cause: Other | 42
  Number of Deaths by Cause: Adverse Event (Total) | 35
  Infections and Infestations (SOC) | 11
  Peritonitis (PT) | 1
  Pneumonia (PT) | 5
  Respiratory Tract Infection (PT) | 1
  Sepsis (PT) | 3
  Septic Shock (PT) | 1
  Cardiac Disorders (SOC) | 7
  Cardiac Arrest (PT) | 2
  Cardiac Failure (PT) | 1
  Cardiac Failure Congestive (PT) | 1
  Cardio-respiratory Arrest (PT) | 1
  Myocardial Infarction (PT) | 1
  Right Ventricular Failure (PT) | 1
  General Disorders & Admin. Site Conditions (SOC) | 6
  Death (PT) | 6
  Blood and Lymphatic System Disorders (SOC) | 3
  Febrile Neutropenia (PT) | 1
  Neutropenia (PT) | 1
  Thrombocytopenia (PT) | 1
  Respiratory, Thoracic & Mediast. Disorders (SOC) | 3
  Acute Respiratory Distress Syndrome (PT) | 1
  Aspiration (PT) | 1
  Pneumonitis (PT) | 1
  Gastrointestinal Disorders (SOC) | 2
  Pancreatitis (PT) | 1
  Pancreatitis Chronic (PT) | 1
  Nervous System Disorders (SOC) | 2
  Hepatic Encephalopathy (PT) | 1
  Ischemic Stroke (PT) | 1
  Metabolism and Nutrition Disorders (SOC) | 1
  Hypoglycaemia (PT) | 1
  Hepatobiliary Disorders (SOC) | 1
  Hepatic Failure (PT) | 1
  Psychiatric Disorders (SOC) | 1
  Delirium (PT) | 1

3. Primary Outcome: Number of Participants Who Died Within 6 Months of Starting Study Treatment by Reported Cause of Death (Adverse Events Leading to Death by System Organ Class and Preferred Term)
Description: as for outcome 2
Time Frame: The median (full range) duration of follow-up was 68.73 (0.03-87.29) months.
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Total Number of Deaths | 38
  Number of Deaths by Cause: Progressive Disease | 18
  Number of Deaths by Cause: Other | 1
  Number of Deaths by Cause: Adverse Event (Total) | 19
  Infections and Infestations (SOC) | 6
  Peritonitis (PT) | 1
  Pneumonia (PT) | 2
  Respiratory Tract Infection (PT) | 1
  Sepsis (PT) | 2
  General Disorders & Admin. Site Conditions (SOC) | 4
  Death (PT) | 4
  Blood and Lymphatic System Disorders (SOC) | 3
  Febrile Neutropenia (PT) | 1
  Neutropenia (PT) | 1
  Thrombocytopenia (PT) | 1
  Cardiac Disorders (SOC) | 2
  Cardiac Arrest (PT) | 1
  Cardio-Respiratory Arrest (PT) | 1
  Respiratory, Thoracic & Mediast. Disorders (SOC) | 2
  Acute Respiratory Distress Syndrome (PT) | 1
  Pneumonitis (PT) | 1
  Gastrointestinal Disorders (SOC) | 1
  Pancreatitis (PT) | 1
  Nervous System Disorders (SOC) | 1
  Hepatic Encephalopathy (PT) | 1
  Metabolism and Nutrition Disorders (SOC) | 1
  Hypoglycaemia (PT) | 1
  Hepatobiliary Disorders (SOC) | 1
  Hepatic Failure (PT) | 1

4. Primary Outcome: Number of Participants With Grade ≥3 Treatment-Emergent Adverse Events, Occurring in ≥1% of Participants by System Organ Class and Preferred Term
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. MedDRA version 22.1 was used to code AEs by system organ class (SOC) and preferred term (PT); PTs that are part of a given SOC are listed in the rows directly below each SOC within the results table. If a participant experienced the same AE at more than one severity grade, only the most severe grade was presented.
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any TEAE - Grade (Gr.) 3 | 676
  Any TEAE - Gr. 4 | 172
  Any TEAE - Gr. 5 | 31
  Gastrointestinal Disorders (SOC) - Gr. 3 | 163
  Gastrointestinal Disorders (SOC) - Gr. 4 | 4
  Gastrointestinal Disorders (SOC) - Gr. 5 | 2
  Diarrhoea (PT) - Gr. 3 | 119
  Diarrhoea (PT) - Gr. 4 | 1
  Diarrhoea (PT) - Gr. 5 | 0
  Vomiting (PT) - Gr. 3 | 19
  Vomiting (PT) - Gr. 4 | 0
  Vomiting (PT) - Gr. 5 | 0
  Skin & Subcutaneous Tissue Disorders (SOC) - Gr. 3 | 56
  Skin & Subcutaneous Tissue Disorders (SOC) - Gr. 4 | 0
  Skin & Subcutaneous Tissue Disorders (SOC) - Gr. 5 | 0
  Gen. Disorders & Admin.Site Conditions (SOC)-Gr. 3 | 100
  Gen. Disorders & Admin.Site Conditions (SOC)-Gr. 4 | 0
  Gen. Disorders & Admin.Site Conditions (SOC)-Gr. 5 | 3
  Fatigue (PT) - Gr. 3 | 36
  Fatigue (PT) - Gr. 4 | 0
  Fatigue (PT) - Gr. 5 | 0
  Asthenia (PT) - Gr. 3 | 29
  Asthenia (PT) - Gr. 4 | 0
  Asthenia (PT) - Gr. 5 | 0
  Mucosal Inflammation (PT) - Gr. 3 | 14
  Mucosal Inflammation (PT) - Gr. 4 | 0
  Mucosal Inflammation (PT) - Gr. 5 | 0
  Nervous System Disorders (SOC) - Gr. 3 | 139
  Nervous System Disorders (SOC) - Gr. 4 | 0
  Nervous System Disorders (SOC) - Gr. 5 | 2
  Neuropathy Peripheral (PT) - Gr. 3 | 26
  Neuropathy Peripheral (PT) - Gr. 4 | 0
  Neuropathy Peripheral (PT) - Gr. 5 | 0
  Syncope (PT) - Gr. 3 | 24
  Syncope (PT) - Gr. 4 | 0
  Syncope (PT) - Gr. 5 | 0
  Headache (PT) - Gr. 3 | 17
  Headache (PT) - Gr. 4 | 0
  Headache (PT) - Gr. 5 | 0
  Paraesthesia (PT) - Gr. 3 | 14
  Paraesthesia (PT) - Gr. 4 | 0
  Paraesthesia (PT) - Gr. 5 | 0
  Peripheral Sensory Neuropathy (PT) - Gr. 3 | 14
  Peripheral Sensory Neuropathy (PT) - Gr. 4 | 0
  Peripheral Sensory Neuropathy (PT) - Gr. 5 | 0
  Infections and Infestations (SOC) - Gr. 3 | 148
  Infections and Infestations (SOC) - Gr. 4 | 19
  Infections and Infestations (SOC) - Gr. 5 | 10
  Pneumonia (PT) - Gr. 3 | 22
  Pneumonia (PT) - Gr. 4 | 1
  Pneumonia (PT) - Gr. 5 | 4
  Vascular Device Infection (PT) - Gr. 3 | 14
  Vascular Device Infection (PT) - Gr. 4 | 0
  Vascular Device Infection (PT) - Gr. 5 | 0
  Device Related Infection (PT) - Gr. 3 | 14
  Device Related Infection (PT) - Gr. 4 | 0
  Device Related Infection (PT) - Gr. 5 | 0
  Musculo. & Connective Tissue Disorders (SOC)-Gr. 3 | 75
  Musculo. & Connective Tissue Disorders (SOC)-Gr. 4 | 0
  Musculo. & Connective Tissue Disorders (SOC)-Gr. 5 | 0
  Resp., Thoracic & Mediast. Disorders (SOC) - Gr. 3 | 62
  Resp., Thoracic & Mediast. Disorders (SOC) - Gr. 4 | 5
  Resp., Thoracic & Mediast. Disorders (SOC) - Gr. 5 | 3
  Pulmonary Embolism (PT) - Gr. 3 | 21
  Pulmonary Embolism (PT) - Gr. 4 | 2
  Pulmonary Embolism (PT) - Gr. 5 | 0
  Dyspnoea (PT) - Gr. 3 | 19
  Dyspnoea (PT) - Gr. 4 | 1
  Dyspnoea (PT) - Gr. 5 | 0
  Blood & Lymphatic System Disorders (SOC) - Gr. 3 | 158
  Blood & Lymphatic System Disorders (SOC) - Gr. 4 | 104
  Blood & Lymphatic System Disorders (SOC) - Gr. 5 | 3
  Neutropenia (PT) - Gr. 3 | 77
  Neutropenia (PT) - Gr. 4 | 67
  Neutropenia (PT) - Gr. 5 | 1
  Febrile Neutropenia (PT) - Gr. 3 | 51
  Febrile Neutropenia (PT) - Gr. 4 | 38
  Febrile Neutropenia (PT) - Gr. 5 | 1
  Anaemia (PT) - Gr. 3 | 29
  Anaemia (PT) - Gr. 4 | 0
  Anaemia (PT) - Gr. 5 | 0
  Leukopenia (PT) - Gr. 3 | 15
  Leukopenia (PT) - Gr. 4 | 3
  Leukopenia (PT) - Gr. 5 | 0
  Investigations (SOC) - Gr. 3 | 116
  Investigations (SOC) - Gr. 4 | 20
  Investigations (SOC) - Gr. 5 | 0
  Neutrophil Count Decreased (PT) - Gr. 3 | 25
  Neutrophil Count Decreased (PT) - Gr. 4 | 13
  Neutrophil Count Decreased (PT) - Gr. 5 | 0
  Ejection Fraction Decreased (PT) - Gr. 3 | 22
  Ejection Fraction Decreased (PT) - Gr. 4 | 2
  Ejection Fraction Decreased (PT) - Gr. 5 | 0
  Gamma-Glutamyltransferase Increased (PT) - Gr. 3 | 19
  Gamma-Glutamyltransferase Increased (PT) - Gr. 4 | 1
  Gamma-Glutamyltransferase Increased (PT) - Gr. 5 | 0
  White Blood Cell Count Decreased (PT) - Gr. 3 | 16
  White Blood Cell Count Decreased (PT) - Gr. 4 | 2
  White Blood Cell Count Decreased (PT) - Gr. 5 | 0
  Alanine Aminotransferase Increased (PT) - Gr. 3 | 16
  Alanine Aminotransferase Increased (PT) - Gr. 4 | 0
  Alanine Aminotransferase Increased (PT) - Gr. 5 | 0
  Metabolism and Nutrition Disorders (SOC) - Gr. 3 | 63
  Metabolism and Nutrition Disorders (SOC) - Gr. 4 | 8
  Metabolism and Nutrition Disorders (SOC) - Gr. 5 | 1
  Hypokalaemia (PT) - Gr. 3 | 19
  Hypokalaemia (PT) - Gr. 4 | 1
  Hypokalaemia (PT) - Gr. 5 | 0
  Vascular Disorders (SOC) - Gr. 3 | 62
  Vascular Disorders (SOC) - Gr. 4 | 2
  Vascular Disorders (SOC) - Gr. 5 | 0
  Hypertension (PT) - Gr. 3 | 45
  Hypertension (PT) - Gr. 4 | 1
  Hypertension (PT) - Gr. 5 | 0
  Psychiatric Disorders (SOC) - Gr. 3 | 15
  Psychiatric Disorders (SOC) - Gr. 4 | 3
  Psychiatric Disorders (SOC) - Gr. 5 | 1
  Injury, Poisoning & Proced. Complicat. (SOC)-Gr. 3 | 43
  Injury, Poisoning & Proced. Complicat. (SOC)-Gr. 4 | 6
  Injury, Poisoning & Proced. Complicat. (SOC)-Gr. 5 | 0
  Cardiac Disorders (SOC) - Gr. 3 | 35
  Cardiac Disorders (SOC) - Gr. 4 | 5
  Cardiac Disorders (SOC) - Gr. 5 | 7
  Immune System Disorders (SOC) - Gr. 3 | 17
  Immune System Disorders (SOC) - Gr. 4 | 1
  Immune System Disorders (SOC) - Gr. 5 | 0
  Renal and Urinary Disorders (SOC) - Gr. 3 | 15
  Renal and Urinary Disorders (SOC) - Gr. 4 | 3
  Renal and Urinary Disorders (SOC) - Gr. 5 | 0
  Neoplasms Benign, Malignant & Unspec. (SOC) -Gr. 3 | 13
  Neoplasms Benign, Malignant & Unspec. (SOC) -Gr. 4 | 5
  Neoplasms Benign, Malignant & Unspec. (SOC) -Gr. 5 | 0
  Hepatobiliary Disorders (SOC) - Gr. 3 | 13
  Hepatobiliary Disorders (SOC) - Gr. 4 | 0
  Hepatobiliary Disorders (SOC) - Gr. 5 | 1

5. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events of Any Grade That Were Related to Study Treatment (Pertuzumab, Trastuzumab, or Taxane), Occurring in ≥10% of Participants by System Organ Class
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. MedDRA version 22.1 was used to code AEs and the system organ classes are presented in descending order according to the total frequency of occurrence. If a participant experienced more than one event in a category, they were counted only once in that category.
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any TEAE Related to Pertuzumab (Rel to Ptz) | 1037
  Rel to Ptz: Gastrointestinal Disorders | 629
  Rel to Ptz: Skin and Subcutaneous Tissue Disorders | 491
  Rel to Ptz: Gen. Disorders & Admin.Site Conditions | 462
  Rel to Ptz: Investigations | 252
  Rel to Ptz: Nervous System Disorders | 207
  Rel to Ptz: Resp., Thoracic & Mediast. Disorders | 188
  Rel to Ptz: Musculo. & Connective Tissue Disorders | 184
  Rel to Ptz: Blood & Lymphatic System Disorders | 182
  Rel to Ptz: Infections and Infestations | 151
  Any TEAE Related to Trastuzumab (Rel to Trz) | 946
  Rel to Trz: Gastrointestinal Disorders | 435
  Rel to Trz: Gen. Disorders & Admin.Site Conditions | 434
  Rel to Trz: Skin and Subcutaneous Tissue Disorders | 384
  Rel to Trz: Investigations | 262
  Rel to Trz: Nervous System Disorders | 184
  Rel to Trz: Musculo. & Connective Tissue Disorders | 179
  Rel to Trz: Blood & Lymphatic System Disorders | 163
  Rel to Trz: Resp., Thoracic & Mediast. Disorders | 153
  Any TEAE Related to Taxane (Rel to Tax) | 1342
  Rel to Tax: Gastrointestinal Disorders | 984
  Rel to Tax: Skin and Subcutaneous Tissue Disorders | 938
  Rel to Tax: Gen. Disorders & Admin.Site Conditions | 834
  Rel to Tax: Nervous System Disorders | 764
  Rel to Tax: Blood & Lymphatic System Disorders | 457
  Rel to Tax: Musculo. & Connective Tissue Disorders | 386
  Rel to Tax: Infections and Infestations | 293
  Rel to Tax: Resp., Thoracic & Mediast. Disorders | 290
  Rel to Tax: Metabolism and Nutrition Disorders | 227
  Rel to Tax: Investigations | 201
  Rel to Tax: Eye Disorders | 174

6. Primary Outcome: Number of Participants With Grade ≥3 Treatment-Emergent Adverse Events That Were Related to Study Treatment (Pertuzumab, Trastuzumab, or Taxane), Occurring in ≥0.5% of Participants by Preferred Term
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. MedDRA version 22.1 was used to code AEs and the preferred terms are presented in descending order according to the total frequency of occurrence. If a participant experienced more than one event in a category, they were counted only once in that category.
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any Grade ≥3 TEAE Related to Pertuz. (Rel to Ptz) | 286
  Rel to Ptz: Diarrhoea | 59
  Rel to Ptz: Neutropenia | 28
  Rel to Ptz: Febrile Neutropenia | 28
  Rel to Ptz: Ejection Fraction Decreased | 19
  Rel to Ptz: Neutrophil Count Decreased | 15
  Rel to Ptz: Fatigue | 15
  Rel to Ptz: Left Ventricular Dysfunction | 10
  Rel to Ptz: Asthenia | 10
  Rel to Ptz: White Blood Cell Count Decreased | 10
  Rel to Ptz: Cardiac Failure | 9
  Any Grade ≥3 TEAE Related to Trastuz. (Rel to Trz) | 245
  Rel to Trz: Diarrhoea | 32
  Rel to Trz: Neutropenia | 30
  Rel to Trz: Ejection Fraction Decreased | 23
  Rel to Trz: Febrile Neutropenia | 21
  Rel to Trz: Neutrophil Count Decreased | 15
  Rel to Trz: Fatigue | 14
  Rel to Trz: Left Ventricular Dysfunction | 11
  Rel to Trz: White Blood Cell Count Decreased | 10
  Rel to Trz: Cardiac Failure | 8
  Rel to Trz: Asthenia | 8
  Any Grade ≥3 TEAE Related to Taxane (Rel to Tax) | 514
  Rel to Tax: Neutropenia | 140
  Rel to Tax: Febrile Neutropenia | 86
  Rel to Tax: Diarrhoea | 80
  Rel to Tax: Neutrophil Count Decreased | 34
  Rel to Tax: Fatigue | 26
  Rel to Tax: Peripheral Neuropathy | 24
  Rel to Tax: Asthenia | 20
  Rel to Tax: Leukopenia | 16
  Rel to Tax: White Blood Cell Count Decreased | 16
  Rel to Tax: Mucosal Inflammation | 14
  Rel to Tax: Paraesthesia | 13
  Rel to Tax: Peripheral Sensory Neuropathy | 13
  Rel to Tax: Onycholysis | 10
  Rel to Tax: Neutropenic Sepsis | 10
  Rel to Tax: Anaemia | 10
  Rel to Tax: Vomiting | 7
  Rel to Tax: Neurotoxicity | 7

7. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events Leading to Discontinuation of Study Treatment (Pertuzumab, Trastuzumab, or Taxane), Occurring in ≥0.2% of Participants by Preferred Term
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. MedDRA version 22.1 was used to code AEs and the preferred terms are presented in descending order according to the total frequency of occurrence. If a participant experienced more than one event in a category, they were counted only once in that category. Discont. = discontinuation; Ptz = pertuzumab; Tax = taxane; Trz = trastuzumab
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any TEAE, Pertuzumab Discontinuation (Ptz Discont) | 140
  Ptz Discont: Ejection Fraction Decreased | 37
  Ptz Discont: Cardiac Failure | 10
  Ptz Discont: Left Ventricular Dysfunction | 7
  Ptz Discont: Diarrhoea | 7
  Ptz Discont: Dyspnoea | 4
  Ptz Discont: Infusion Related Reaction | 4
  Ptz Discont: Sepsis | 3
  Ptz Discont: Neuropathy Peripheral | 3
  Ptz Discont: Hypersensitivity | 3
  Ptz Discont: General Physical Health Deterioration | 3
  Any TEAE, Trastuzumab Discontinuation(Trz Discont) | 133
  Trz Discont: Ejection Fraction Decreased | 37
  Trz Discont: Cardiac Failure | 10
  Trz Discont: Left Ventricular Dysfunction | 7
  Trz Discont: Diarrhoea | 6
  Trz Discont: Sepsis | 3
  Trz Discont: Dyspnoea | 3
  Trz Discont: Neuropathy Peripheral | 3
  Trz Discont: Hypersensitivity | 3
  Trz Discont: General Physical Health Deterioration | 3
  Any TEAE, Taxane Discontinuation (Tax Discont) | 286
  Tax Discont: Neuropathy Peripheral | 52
  Tax Discont: Peripheral Sensory Neuropathy | 25
  Tax Discont: Paraesthesia | 24
  Tax Discont: Diarrhoea | 19
  Tax Discont: Fatigue | 16
  Tax Discont: Asthenia | 13
  Tax Discont: Onycholysis | 8
  Tax Discont: Nail Toxicity | 7
  Tax Discont: Neurotoxicity | 7
  Tax Discont: Polyneuropathy | 7
  Tax Discont: Oedema Peripheral | 7
  Tax Discont: Febrile Neutropenia | 7
  Tax Discont: Neutropenia | 7
  Tax Discont: Dyspnoea | 6
  Tax Discont: Decreased Appetite | 6
  Tax Discont: Ejection Fraction Decreased | 5
  Tax Discont: General Physical Health Deterioration | 4
  Tax Discont: Mucosal Inflammation | 4
  Tax Discont: Rash | 4
  Tax Discont: Anaemia | 4
  Tax Discont: Arthralgia | 4
  Tax Discont: Drug Hypersensitivity | 4
  Tax Discont: Dysgeusia | 3
  Tax Discont: Nail Disorder | 3
  Tax Discont: Nail Dystrophy | 3
  Tax Discont: Skin Toxicity | 3
  Tax Discont: Pneumonia | 3
  Tax Discont: Sepsis | 3
  Tax Discont: Pleural Effusion | 3
  Tax Discont: Pneumonitis | 3
  Tax Discont: Cardiac Failure | 3
  Tax Discont: Myalgia | 3

8. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events Leading to Dose Interruption of Study Treatment (Pertuzumab, Trastuzumab, or Taxane), Occurring in ≥0.5% of Participants by Preferred Term
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. MedDRA version 22.1 was used to code AEs and the preferred terms are presented in descending order according to the total frequency of occurrence. If a participant experienced more than one event in a category, they were counted only once in that category. Interrupt. = interruption; Ptz = pertuzumab; Tax = taxane; Trz = trastuzumab
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any TEAE, Pertuzumab Interruption (Ptz Interrupt) | 334
  Ptz Interrupt: Ejection Fraction Decreased | 51
  Ptz Interrupt: Diarrhoea | 21
  Ptz Interrupt: Neutropenia | 17
  Ptz Interrupt: Pneumonia | 14
  Ptz Interrupt: Upper Respiratory Tract Infection | 13
  Ptz Interrupt: Pyrexia | 11
  Ptz Interrupt: Dyspnoea | 11
  Ptz Interrupt: Drug Hypersensitivity | 9
  Ptz Interrupt: Influenza | 8
  Ptz Interrupt: Asthenia | 8
  Ptz Interrupt: Neutrophil Count Decreased | 8
  Ptz Interrupt: Nasopharyngitis | 7
  Ptz Interrupt: Anaemia | 7
  Any TEAE, Trastuzumab Interruption (Trz Interrupt) | 386
  Trz Interrupt: Ejection Fraction Decreased | 52
  Trz Interrupt: Drug Hypersensitivity | 31
  Trz Interrupt: Diarrhoea | 20
  Trz Interrupt: Pyrexia | 18
  Trz Interrupt: Neutropenia | 17
  Trz Interrupt: Dyspnoea | 17
  Trz Interrupt: Pneumonia | 14
  Trz Interrupt: Chills | 13
  Trz Interrupt: Infusion Related Reaction | 13
  Trz Interrupt: Upper Respiratory Tract Infection | 12
  Trz Interrupt: Neutrophil Count Decreased | 8
  Trz Interrupt: Influenza | 7
  Trz Interrupt: Asthenia | 7
  Trz Interrupt: Vomiting | 7
  Trz Interrupt: Anaemia | 7
  Trz Interrupt: Nasopharyngitis | 7
  Any TEAE, Taxane Interruption (Tax Interrupt) | 354
  Tax Interrupt: Neutropenia | 46
  Tax Interrupt: Diarrhoea | 30
  Tax Interrupt: Leukopenia | 17
  Tax Interrupt: Dyspnoea | 15
  Tax Interrupt: Pyrexia | 14
  Tax Interrupt: Neutrophil Count Decreased | 14
  Tax Interrupt: Ejection Fraction Decreased | 13
  Tax Interrupt: Neuropathy Peripheral | 13
  Tax Interrupt: Nasopharyngitis | 10
  Tax Interrupt: Drug Hypersensitivity | 10
  Tax Interrupt: Fatigue | 10
  Tax Interrupt: Upper Respiratory Tract Infection | 9
  Tax Interrupt: Infusion Related Reaction | 9
  Tax Interrupt: Asthenia | 9
  Tax Interrupt: Erythema | 8
  Tax Interrupt: Pneumonia | 7
  Tax Interrupt: Flushing | 7
  Tax Interrupt: Hypersensitivity | 7

9. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events to Monitor of Any Grade, Occurring in ≥5% of Participants by Category
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first dose of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, it was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. If a participant had more than one event in a category, they were counted only once in that category. TEAEs to monitor included anaphylaxis and hypersensitivity, cardiac dysfunction, diarrhoea Grade ≥3, pregnancy-related AEs, interstitial lung disease, infusion-/administration-related reactions, mucositis, (febrile) neutropenia, rash/skin reactions, and suspected transmission of infectious agent. MedDRA version 22.1 was used to code AEs; AEs may fall within multiple categories.
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any TEAE to Monitor | 1320
  Infusion-/Administration-Related Reactions | 1096
  Rash/Skin Reactions | 668
  Mucositis | 618
  Cardiac Dysfunction | 478
  Neutropenia/Febrile Neutropenia | 439
  Anaphylaxis and Hypersensitivity | 124
  Diarrhoea Grade ≥3 | 120

10. Primary Outcome: Number of Participants With Grade ≥3 Treatment-Emergent Adverse Events to Monitor, Occurring in ≥0.5% of Participants by Category and Preferred Term
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first dose of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, it was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. If a participant had more than one event in a category, they were counted only once in that category. TEAEs to monitor included anaphylaxis and hypersensitivity, cardiac dysfunction, diarrhoea Grade ≥3, pregnancy-related AEs, interstitial lung disease, infusion-/administration-related reactions, mucositis, (febrile) neutropenia, rash/skin reactions, and suspected transmission of infectious agent. MedDRA version 22.1 was used to code AEs; preferred terms (PT) that are part of a given category are listed in the rows directly below each category within the results table.
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any Grade ≥3 TEAE to Monitor | 535
  Neutropenia/Febrile Neutropenia (Category) | 279
  Neutropenia (PT) | 145
  Febrile Neutropenia (PT) | 90
  Neutrophil Count Decreased (PT) | 38
  Leukopenia (PT) | 18
  White Blood Cell Count Decreased (PT) | 18
  Neutropenic Sepsis (PT) | 10
  Infusion-/Admin.-Related Reactions (Category) | 123
  Hypertension (PT) | 27
  IRR/ARR: Drug Hypersensitivity (PT) | 12
  Asthenia (PT) | 11
  Fatigue (PT) | 11
  Dyspnoea (PT) | 10
  Infusion Related Reaction (PT) | 8
  Paraesthesia (PT) | 7
  Diarrhoea Grade ≥3 (Category) | 120
  Diarrhoea (PT) | 120
  Cardiac Dysfunction (Category) | 51
  Ejection Fraction Decreased (PT) | 24
  Left Ventricular Dysfunction (PT) | 11
  Cardiac Failure (PT) | 9
  Mucositis (Category) | 33
  Mucosal Inflammation (PT) | 14
  Stomatitis (PT) | 9
  Rash/Skin Reactions (Category) | 28
  Rash (PT) | 10
  Anaphylaxis and Hypersensitivity (Category) | 18
  Anaphyl./Hypersens.: Drug Hypersensitivity (PT) | 13

11. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events of Special Interest by Category and Preferred Term
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. TEAEs of special interest included LVEF decreased, liver enzymes (ALT or AST) increased, and suspected transmission of infectious agent by the study drug. MedDRA version 22.1 was used to code AEs; preferred terms (PT) that are part of a given category are listed in the rows directly below each category within the results table. If a participant experienced more than one event in a category, they were counted only once in that category.
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Any TEAE of Special Interest | 91
  Decline in LVEF (Category) | 90
  Ejection Fraction Decreased (PT) | 75
  Left Ventricular Dysfunction (PT) | 8
  Cardiac Failure (PT) | 7
  Cardiac Failure Congestive (PT) | 1
  Elevated ALT or AST (Category) | 1
  Hepatic Failure (PT) | 1

12. Primary Outcome: Subgroup Analysis by Region of Enrollment: Overview of the Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), Grade ≥3 TEAEs, and Grade ≥3 TEAEs Related to Pertuzumab
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE.
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Europe; Asia; North America; South America; Africa; Other (Australia): Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Taxane chemotherapy was docetaxel, paclitaxel, or nab-paclitaxel, per the investigator's choice.
Arm/Group | Europe | Asia | North America | South America | Africa | Other (Australia)
Number analyzed (Participants) | 1009 | 177 | 34 | 121 | 71 | 24
Participants
  Any Serious TEAE | 385 | 74 | 9 | 37 | 16 | 14
  Any TEAE - Grade 3 or Higher (≥3) | 632 | 109 | 22 | 63 | 37 | 16
  Any Grade ≥3 TEAE Related to Pertuzumab | 187 | 44 | 5 | 27 | 19 | 4

13. Primary Outcome: Subgroup Analysis by Age (≤65 vs. >65 Years): Overview of the Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), TEAEs Leading to Death, Grade ≥3 TEAEs, Any-Grade and Grade ≥3 TEAEs Related to Pertuzumab, and TEAEs to Monitor
Description: Treatment-emergent adverse events (TEAEs) were adverse events (AEs) that started or worsened in severity on or after the first administration of study drug, up to and including 28 days after the last dose. The investigator graded all AEs for severity per NCI-CTCAE v4.0; if not listed, the AE was assessed as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening/disabling; Grade 5 = death. The investigator determined whether an AE was related to study drug and independently assessed severity and seriousness of each AE. TEAEs to monitor included anaphylaxis and hypersensitivity, cardiac dysfunction, diarrhoea Grade ≥3, pregnancy-related AEs, interstitial lung disease, infusion-/administration-related reactions, mucositis, (febrile) neutropenia, rash/skin reactions, and suspected transmission of infectious agent.
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Age ≤65 Years; Age >65 Years: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Taxane chemotherapy was docetaxel, paclitaxel, or nab-paclitaxel, per the investigator's choice.
Arm/Group | Age ≤65 Years | Age >65 Years
Number analyzed (Participants) | 1167 | 269
Participants
  Any Serious TEAE | 415 | 120
  Any TEAE Leading to Death | 17 | 14
  Any TEAE - Grade 3 or Higher (≥3) | 688 | 191
  Any TEAE Related to Pertuzumab - Any Grade | 845 | 192
  Any Grade ≥3 TEAE Related to Pertuzumab | 224 | 62
  Any TEAE to Monitor - Any Grade | 1081 | 239

14. Primary Outcome: Subgroup Analysis by Taxane Chemotherapy: Overview of the Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), TEAEs Leading to Death, Grade ≥3 TEAEs, Any-Grade and Grade ≥3 TEAEs Related to Pertuzumab, and TEAEs to Monitor
Description: as for outcome 13
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment. Only participants who received any taxane chemotherapy during the study were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Docetaxel: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Participants in this subgroup received docetaxel as their taxane chemotherapy, per the investigator's choice.
- Paclitaxel: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Participants in this subgroup received paclitaxel as their taxane chemotherapy, per the investigator's choice.
- Nab-Paclitaxel: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Participants in this subgroup received nab-paclitaxel as their taxane chemotherapy, per the investigator's choice.
Arm/Group | Docetaxel | Paclitaxel | Nab-Paclitaxel
Number analyzed (Participants) | 775 | 588 | 65
Participants
  Any Serious TEAE | 300 | 210 | 22
  Any TEAE Leading to Death | 14 | 16 | 1
  Any TEAE - Grade 3 or Higher (≥3) | 491 | 349 | 36
  Any TEAE Related to Pertuzumab - Any Grade | 547 | 434 | 52
  Any Grade ≥3 TEAE Related to Pertuzumab | 171 | 105 | 9
  Any TEAE to Monitor - Any Grade | 709 | 541 | 64

15. Primary Outcome: Subgroup Analysis by ECOG Performance Status at Baseline: Overview of the Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), Grade ≥3 TEAEs, and Grade ≥3 TEAEs Related to Pertuzumab
Description: as for outcome 12
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment. There were 2 participants with missing evaluations for ECOG performance status at baseline who were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- ECOG Performance Status 0 or 1; ECOG Performance Status 2: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Taxane chemotherapy was docetaxel, paclitaxel, or nab-paclitaxel, per the investigator's choice.
Arm/Group | ECOG Performance Status 0 or 1 | ECOG Performance Status 2
Number analyzed (Participants) | 1371 | 63
Participants
  Any Serious TEAE | 502 | 33
  Any TEAE - Grade 3 or Higher (≥3) | 837 | 41
  Any Grade ≥3 TEAE Related to Pertuzumab | 273 | 13

16. Primary Outcome: Subgroup Analysis by Visceral Disease at Baseline: Overview of the Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), Grade ≥3 TEAEs, and Grade ≥3 TEAEs Related to Pertuzumab
Description: as for outcome 12
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Visceral Disease; Non-Visceral Disease: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Taxane chemotherapy was docetaxel, paclitaxel, or nab-paclitaxel, per the investigator's choice.
Arm/Group | Visceral Disease | Non-Visceral Disease
Number analyzed (Participants) | 992 | 444
Participants
  Any Serious TEAE | 353 | 182
  Any TEAE - Grade 3 or Higher (≥3) | 610 | 269
  Any Grade ≥3 TEAE Related to Pertuzumab | 197 | 89

17. Primary Outcome: Subgroup Analysis by Prior (Neo)Adjuvant Chemotherapy: Overview of the Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), Grade ≥3 TEAEs, and Grade ≥3 TEAEs Related to Pertuzumab
Description: as for outcome 12
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Prior (Neo)Adjuvant Chemotherapy; No Prior (Neo)Adjuvant Chemotherapy: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Taxane chemotherapy was docetaxel, paclitaxel, or nab-paclitaxel, per the investigator's choice.
Arm/Group | Prior (Neo)Adjuvant Chemotherapy | No Prior (Neo)Adjuvant Chemotherapy
Number analyzed (Participants) | 786 | 650
Participants
  Any Serious TEAE | 283 | 252
  Any TEAE - Grade 3 or Higher (≥3) | 493 | 386
  Any Grade ≥3 TEAE Related to Pertuzumab | 169 | 117

18. Primary Outcome: Subgroup Analysis by Hormone Receptor Status at Baseline: Overview of the Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), Grade ≥3 TEAEs, and Grade ≥3 TEAEs Related to Pertuzumab
Description: as for outcome 12
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Hormone Receptor Positive; Hormone Receptor Negative; Hormone Receptor Status Unknown: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Taxane chemotherapy was docetaxel, paclitaxel, or nab-paclitaxel, per the investigator's choice.
Arm/Group | Hormone Receptor Positive | Hormone Receptor Negative | Hormone Receptor Status Unknown
Number analyzed (Participants) | 918 | 512 | 6
Participants
  Any Serious TEAE | 353 | 179 | 3
  Any TEAE - Grade 3 or Higher (≥3) | 573 | 303 | 3
  Any Grade ≥3 TEAE Related to Pertuzumab | 181 | 103 | 2

19. Primary Outcome: Subgroup Analysis by Previous Trastuzumab Therapy: Overview of the Number of Participants With Serious Treatment-Emergent Adverse Events (TEAEs), Grade ≥3 TEAEs, and Grade ≥3 TEAEs Related to Pertuzumab
Description: as for outcome 12
Time Frame: as for outcome 1
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Previous Trastuzumab Therapy; No Previous Trastuzumab Therapy: Participants received pertuzumab and trastuzumab intravenously (IV) plus taxane chemotherapy once of every 3 weeks per treatment cycle until predefined study end, unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurred first. Taxane chemotherapy was docetaxel, paclitaxel, or nab-paclitaxel, per the investigator's choice.
Arm/Group | Previous Trastuzumab Therapy | No Previous Trastuzumab Therapy
Number analyzed (Participants) | 400 | 1036
Participants
  Any Serious TEAE | 135 | 400
  Any TEAE - Grade 3 or Higher (≥3) | 238 | 641
  Any Grade ≥3 TEAE Related to Pertuzumab | 77 | 209

20. Primary Outcome: Number of Participants With a Congestive Heart Failure Event
Description: Congestive heart failure was defined as the Standardised MedDRA Query (SMQ) 'Cardiac failure (wide)' from the Medical Dictionary for Regulatory Activities, version 22.1 (MedDRA version 22.1).
Time Frame: From Baseline until 28 days after the last dose of study treatment. The median (full range) duration of exposure to any study treatment was 16.2 (0.0-86.4) months.
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants | 478

21. Primary Outcome: Time to Onset of the First Episode of Congestive Heart Failure
Description: Congestive heart failure was defined as SMQ 'Cardiac failure (wide)' from the MedDRA version 22.1. Time to onset of the first episode of congestive heart failure was analyzed using a Kaplan-Meier approach. Participants who did not experience any congestive heart failure at the time of data-cut were censored at the date of the last attended visit whilst on-treatment (including visits up to and including 28 days after last dose of study treatment). Only treatment emergent congestive heart failure events are included.
Time Frame: as for outcome 20
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Months | NA [73.82 to NA] — The median and upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study.

22. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) Values Over the Course of the Study
Description: All participants must have had a baseline LVEF ≥50% to enroll in the study; patients with significant cardiac disease or baseline LVEF below 50% were not eligible for this study. The change from baseline LVEF values were reported at every 3 cycles over the course of the study and at the final treatment, worst treatment, and maximum decrease values. The final treatment value was defined as the last LVEF value observed before all study treatment discontinuation. The worst treatment value was defined as the lowest LVEF value observed before all study treatment discontinuation. The maximum decrease value was defined as the largest decrease of LVEF value from baseline, or minimum increase if a participant's post-baseline LVEF measures were all larger than the baseline value.
Time Frame: Baseline, predose on Day 1 of every 3 cycles (1 cycle is 3 weeks) during treatment period, and 28 days post-treatment safety follow-up. The median (full range) duration of exposure to any study treatment was 16.2 (0.0-86.4) months.
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Mean (Standard Deviation); unit: Percentage points of LVEF
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Percentage points of LVEF
  Baseline (BL): Absolute Value at Visit: number analyzed (Participants) | 1435
  Baseline (BL): Absolute Value at Visit | 64.6 (6.46)
  Change from BL at Cycle 3: number analyzed (Participants) | 1311
  Change from BL at Cycle 3 | -1.1 (6.49)
  Change from BL at Cycle 6: number analyzed (Participants) | 1248
  Change from BL at Cycle 6 | -1.5 (6.60)
  Change from BL at Cycle 9: number analyzed (Participants) | 1150
  Change from BL at Cycle 9 | -2.1 (6.56)
  Change from BL at Cycle 12: number analyzed (Participants) | 1028
  Change from BL at Cycle 12 | -1.9 (6.66)
  Change from BL at Cycle 15: number analyzed (Participants) | 898
  Change from BL at Cycle 15 | -2.2 (6.50)
  Change from BL at Cycle 18: number analyzed (Participants) | 816
  Change from BL at Cycle 18 | -1.8 (6.77)
  Change from BL at Cycle 21: number analyzed (Participants) | 731
  Change from BL at Cycle 21 | -1.9 (6.79)
  Change from BL at Cycle 24: number analyzed (Participants) | 681
  Change from BL at Cycle 24 | -1.9 (6.93)
  Change from BL at Cycle 27: number analyzed (Participants) | 633
  Change from BL at Cycle 27 | -2.1 (6.81)
  Change from BL at Cycle 30: number analyzed (Participants) | 589
  Change from BL at Cycle 30 | -1.8 (6.80)
  Change from BL at Cycle 33: number analyzed (Participants) | 558
  Change from BL at Cycle 33 | -1.9 (6.97)
  Change from BL at Cycle 36: number analyzed (Participants) | 509
  Change from BL at Cycle 36 | -2.1 (6.53)
  Change from BL at Cycle 39: number analyzed (Participants) | 480
  Change from BL at Cycle 39 | -2.1 (6.77)
  Change from BL at Cycle 42: number analyzed (Participants) | 451
  Change from BL at Cycle 42 | -1.9 (6.52)
  Change from BL at Cycle 45: number analyzed (Participants) | 428
  Change from BL at Cycle 45 | -2.2 (6.94)
  Change from BL at Cycle 48: number analyzed (Participants) | 390
  Change from BL at Cycle 48 | -2.1 (6.67)
  Change from BL at Cycle 51: number analyzed (Participants) | 357
  Change from BL at Cycle 51 | -1.6 (6.75)
  Change from BL at Cycle 54: number analyzed (Participants) | 325
  Change from BL at Cycle 54 | -1.7 (6.38)
  Change from BL at Cycle 57: number analyzed (Participants) | 332
  Change from BL at Cycle 57 | -1.7 (6.87)
  Change from BL at Cycle 60: number analyzed (Participants) | 313
  Change from BL at Cycle 60 | -1.5 (6.46)
  Change from BL at Cycle 63: number analyzed (Participants) | 302
  Change from BL at Cycle 63 | -1.6 (7.13)
  Change from BL at Cycle 66: number analyzed (Participants) | 284
  Change from BL at Cycle 66 | -2.0 (6.63)
  Change from BL at Cycle 69: number analyzed (Participants) | 270
  Change from BL at Cycle 69 | -1.9 (6.45)
  Change from BL at Cycle 72: number analyzed (Participants) | 259
  Change from BL at Cycle 72 | -2.1 (6.80)
  Change from BL at Cycle 75: number analyzed (Participants) | 254
  Change from BL at Cycle 75 | -1.5 (6.84)
  Change from BL at Cycle 78: number analyzed (Participants) | 245
  Change from BL at Cycle 78 | -1.8 (7.41)
  Change from BL at Cycle 81: number analyzed (Participants) | 226
  Change from BL at Cycle 81 | -1.8 (6.98)
  Change from BL at Cycle 84: number analyzed (Participants) | 215
  Change from BL at Cycle 84 | -1.6 (6.89)
  Change from BL at Cycle 87: number analyzed (Participants) | 196
  Change from BL at Cycle 87 | -1.9 (6.31)
  Change from BL at Cycle 90: number analyzed (Participants) | 177
  Change from BL at Cycle 90 | -1.1 (6.68)
  Change from BL at Cycle 93: number analyzed (Participants) | 156
  Change from BL at Cycle 93 | -1.6 (6.78)
  Change from BL at Cycle 96: number analyzed (Participants) | 128
  Change from BL at Cycle 96 | -1.8 (6.33)
  Change from BL at Cycle 99: number analyzed (Participants) | 106
  Change from BL at Cycle 99 | -2.0 (7.20)
  Change from BL at Cycle 102: number analyzed (Participants) | 82
  Change from BL at Cycle 102 | -2.5 (7.95)
  Change from BL at Cycle 105: number analyzed (Participants) | 65
  Change from BL at Cycle 105 | -2.5 (6.86)
  Change from BL at Cycle 108: number analyzed (Participants) | 49
  Change from BL at Cycle 108 | -1.8 (8.04)
  Change from BL at Cycle 111: number analyzed (Participants) | 42
  Change from BL at Cycle 111 | -3.3 (7.47)
  Change from BL at Cycle 114: number analyzed (Participants) | 23
  Change from BL at Cycle 114 | -1.1 (8.12)
  Change from BL at Cycle 117: number analyzed (Participants) | 17
  Change from BL at Cycle 117 | -5.8 (7.48)
  Change from BL at Cycle 120: number analyzed (Participants) | 7
  Change from BL at Cycle 120 | -8.6 (6.70)
  Change from BL at Cycle 123: number analyzed (Participants) | 3
  Change from BL at Cycle 123 | -9.3 (3.51)
  Change from BL at Cycle 126: number analyzed (Participants) | 1
  Change from BL at Cycle 126 | -9.0 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at End of Treatment: number analyzed (Participants) | 546
  Change from BL at End of Treatment | -3.8 (8.34)
  Change from BL at Day 28 of Follow-Up: number analyzed (Participants) | 584
  Change from BL at Day 28 of Follow-Up | -3.2 (8.19)
  Change from BL: Final Treatment Value: number analyzed (Participants) | 1360
  Change from BL: Final Treatment Value | -2.0 (6.77)
  Change from BL: Worst Treatment Value: number analyzed (Participants) | 1360
  Change from BL: Worst Treatment Value | -7.1 (6.88)
  Change from BL: Maximum Decrease Value: number analyzed (Participants) | 1398
  Change from BL: Maximum Decrease Value | -7.7 (7.45)

23. Primary Outcome: Number of Participants by Change From Baseline in Left Ventricular Ejection Fraction (LVEF) Categories Over the Course of the Study
Description: All participants must have had a baseline LVEF greater than or equal to (≥)50% to enroll in the study; patients with significant cardiac disease or baseline LVEF below 50% were not eligible for this study. The number of participants are reported according to four change from baseline in LVEF value categories over the course of the study: 1) an increase or decrease from baseline LVEF less than (<)10% points or no change in LVEF; 2) an absolute LVEF value <45% points and a decrease from baseline LVEF ≥10% points to <15% points; 3) an absolute LVEF value <45% points and a decrease from baseline LVEF ≥15% points; or 4) an absolute LVEF value ≥45% points and a decrease from baseline LVEF ≥10% points. BL = baseline; Decr. = decrease; Incr. = increase
Time Frame: as for outcome 22
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Cycle 3: number analyzed (Participants) | 1311
  Cycle 3: Incr. or Decr. from BL <10% Points, or No Change | 1190
  Cycle 3: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 2
  Cycle 3: LVEF<45% Points and Decr. from BL ≥15% Points | 5
  Cycle 3: LVEF≥45% Points and Decr. from BL ≥10% Points | 114
  Cycle 6: number analyzed (Participants) | 1248
  Cycle 6: Incr. or Decr. from BL <10% Points, or No Change | 1110
  Cycle 6: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 6: LVEF<45% Points and Decr. from BL ≥15% Points | 2
  Cycle 6: LVEF≥45% Points and Decr. from BL ≥10% Points | 136
  Cycle 9: number analyzed (Participants) | 1150
  Cycle 9: Incr. or Decr. from BL <10% Points, or No Change | 1005
  Cycle 9: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 2
  Cycle 9: LVEF<45% Points and Decr. from BL ≥15% Points | 4
  Cycle 9: LVEF≥45% Points and Decr. from BL ≥10% Points | 139
  Cycle 12: number analyzed (Participants) | 1028
  Cycle 12: Incr. or Decr. from BL <10% Points, or No Change | 906
  Cycle 12: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 12: LVEF<45% Points and Decr. from BL ≥15% Points | 6
  Cycle 12: LVEF≥45% Points and Decr. from BL ≥10% Points | 116
  Cycle 15: number analyzed (Participants) | 898
  Cycle 15: Incr. or Decr. from BL <10% Points, or No Change | 780
  Cycle 15: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 3
  Cycle 15: LVEF<45% Points and Decr. from BL ≥15% Points | 6
  Cycle 15: LVEF≥45% Points and Decr. from BL ≥10% Points | 109
  Cycle 18: number analyzed (Participants) | 816
  Cycle 18: Incr. or Decr. from BL <10% Points, or No Change | 719
  Cycle 18: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 18: LVEF<45% Points and Decr. from BL ≥15% Points | 5
  Cycle 18: LVEF≥45% Points and Decr. from BL ≥10% Points | 92
  Cycle 21: number analyzed (Participants) | 731
  Cycle 21: Incr. or Decr. from BL <10% Points, or No Change | 639
  Cycle 21: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 21: LVEF<45% Points and Decr. from BL ≥15% Points | 4
  Cycle 21: LVEF≥45% Points and Decr. from BL ≥10% Points | 88
  Cycle 24: number analyzed (Participants) | 681
  Cycle 24: Incr. or Decr. from BL <10% Points, or No Change | 588
  Cycle 24: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 24: LVEF<45% Points and Decr. from BL ≥15% Points | 2
  Cycle 24: LVEF≥45% Points and Decr. from BL ≥10% Points | 91
  Cycle 27: number analyzed (Participants) | 633
  Cycle 27: Incr. or Decr. from BL <10% Points, or No Change | 553
  Cycle 27: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 27: LVEF<45% Points and Decr. from BL ≥15% Points | 2
  Cycle 27: LVEF≥45% Points and Decr. from BL ≥10% Points | 78
  Cycle 30: number analyzed (Participants) | 589
  Cycle 30: Incr. or Decr. from BL <10% Points, or No Change | 518
  Cycle 30: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 30: LVEF<45% Points and Decr. from BL ≥15% Points | 1
  Cycle 30: LVEF≥45% Points and Decr. from BL ≥10% Points | 70
  Cycle 33: number analyzed (Participants) | 558
  Cycle 33: Incr. or Decr. from BL <10% Points, or No Change | 485
  Cycle 33: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 33: LVEF<45% Points and Decr. from BL ≥15% Points | 1
  Cycle 33: LVEF≥45% Points and Decr. from BL ≥10% Points | 72
  Cycle 36: number analyzed (Participants) | 509
  Cycle 36: Incr. or Decr. from BL <10% Points, or No Change | 446
  Cycle 36: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 36: LVEF<45% Points and Decr. from BL ≥15% Points | 1
  Cycle 36: LVEF≥45% Points and Decr. from BL ≥10% Points | 62
  Cycle 39: number analyzed (Participants) | 480
  Cycle 39: Incr. or Decr. from BL <10% Points, or No Change | 414
  Cycle 39: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 1
  Cycle 39: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 39: LVEF≥45% Points and Decr. from BL ≥10% Points | 65
  Cycle 42: number analyzed (Participants) | 451
  Cycle 42: Incr. or Decr. from BL <10% Points, or No Change | 405
  Cycle 42: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 42: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 42: LVEF≥45% Points and Decr. from BL ≥10% Points | 46
  Cycle 45: number analyzed (Participants) | 428
  Cycle 45: Incr. or Decr. from BL <10% Points, or No Change | 358
  Cycle 45: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 45: LVEF<45% Points and Decr. from BL ≥15% Points | 1
  Cycle 45: LVEF≥45% Points and Decr. from BL ≥10% Points | 69
  Cycle 48: number analyzed (Participants) | 390
  Cycle 48: Incr. or Decr. from BL <10% Points, or No Change | 340
  Cycle 48: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 48: LVEF<45% Points and Decr. from BL ≥15% Points | 1
  Cycle 48: LVEF≥45% Points and Decr. from BL ≥10% Points | 49
  Cycle 51: number analyzed (Participants) | 357
  Cycle 51: Incr. or Decr. from BL <10% Points, or No Change | 314
  Cycle 51: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 51: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 51: LVEF≥45% Points and Decr. from BL ≥10% Points | 43
  Cycle 54: number analyzed (Participants) | 325
  Cycle 54: Incr. or Decr. from BL <10% Points, or No Change | 292
  Cycle 54: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 54: LVEF<45% Points and Decr. from BL ≥15% Points | 3
  Cycle 54: LVEF≥45% Points and Decr. from BL ≥10% Points | 30
  Cycle 57: number analyzed (Participants) | 332
  Cycle 57: Incr. or Decr. from BL <10% Points, or No Change | 291
  Cycle 57: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 57: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 57: LVEF≥45% Points and Decr. from BL ≥10% Points | 41
  Cycle 60: number analyzed (Participants) | 313
  Cycle 60: Incr. or Decr. from BL <10% Points, or No Change | 284
  Cycle 60: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 60: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 60: LVEF≥45% Points and Decr. from BL ≥10% Points | 29
  Cycle 63: number analyzed (Participants) | 302
  Cycle 63: Incr. or Decr. from BL <10% Points, or No Change | 263
  Cycle 63: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 63: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 63: LVEF≥45% Points and Decr. from BL ≥10% Points | 39
  Cycle 66: number analyzed (Participants) | 284
  Cycle 66: Incr. or Decr. from BL <10% Points, or No Change | 249
  Cycle 66: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 66: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 66: LVEF≥45% Points and Decr. from BL ≥10% Points | 35
  Cycle 69: number analyzed (Participants) | 270
  Cycle 69: Incr. or Decr. from BL <10% Points, or No Change | 237
  Cycle 69: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 69: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 69: LVEF≥45% Points and Decr. from BL ≥10% Points | 33
  Cycle 72: number analyzed (Participants) | 259
  Cycle 72: Incr. or Decr. from BL <10% Points, or No Change | 224
  Cycle 72: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 72: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 72: LVEF≥45% Points and Decr. from BL ≥10% Points | 35
  Cycle 75: number analyzed (Participants) | 254
  Cycle 75: Incr. or Decr. from BL <10% Points, or No Change | 224
  Cycle 75: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 75: LVEF<45% Points and Decr. from BL ≥15% Points | 1
  Cycle 75: LVEF≥45% Points and Decr. from BL ≥10% Points | 29
  Cycle 78: number analyzed (Participants) | 245
  Cycle 78: Incr. or Decr. from BL <10% Points, or No Change | 214
  Cycle 78: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 78: LVEF<45% Points and Decr. from BL ≥15% Points | 2
  Cycle 78: LVEF≥45% Points and Decr. from BL ≥10% Points | 29
  Cycle 81: number analyzed (Participants) | 226
  Cycle 81: Incr. or Decr. from BL <10% Points, or No Change | 196
  Cycle 81: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 81: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 81: LVEF≥45% Points and Decr. from BL ≥10% Points | 30
  Cycle 84: number analyzed (Participants) | 215
  Cycle 84: Incr. or Decr. from BL <10% Points, or No Change | 192
  Cycle 84: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 84: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 84: LVEF≥45% Points and Decr. from BL ≥10% Points | 23
  Cycle 87: number analyzed (Participants) | 196
  Cycle 87: Incr. or Decr. from BL <10% Points, or No Change | 174
  Cycle 87: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 87: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 87: LVEF≥45% Points and Decr. from BL ≥10% Points | 22
  Cycle 90: number analyzed (Participants) | 177
  Cycle 90: Incr. or Decr. from BL <10% Points, or No Change | 161
  Cycle 90: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 90: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 90: LVEF≥45% Points and Decr. from BL ≥10% Points | 16
  Cycle 93: number analyzed (Participants) | 156
  Cycle 93: Incr. or Decr. from BL <10% Points, or No Change | 140
  Cycle 93: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 93: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 93: LVEF≥45% Points and Decr. from BL ≥10% Points | 16
  Cycle 96: number analyzed (Participants) | 128
  Cycle 96: Incr. or Decr. from BL <10% Points, or No Change | 115
  Cycle 96: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 96: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 96: LVEF≥45% Points and Decr. from BL ≥10% Points | 13
  Cycle 99: number analyzed (Participants) | 106
  Cycle 99: Incr. or Decr. from BL <10% Points, or No Change | 92
  Cycle 99: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 99: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 99: LVEF≥45% Points and Decr. from BL ≥10% Points | 14
  Cycle 102: number analyzed (Participants) | 82
  Cycle 102: Incr. or Decr. from BL <10% Points, or No Change | 68
  Cycle 102: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 102: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 102: LVEF≥45% Points and Decr. from BL ≥10% Points | 14
  Cycle 105: number analyzed (Participants) | 65
  Cycle 105: Incr. or Decr. from BL <10% Points, or No Change | 56
  Cycle 105: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 105: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 105: LVEF≥45% Points and Decr. from BL ≥10% Points | 9
  Cycle 108: number analyzed (Participants) | 49
  Cycle 108: Incr. or Decr. from BL <10% Points, or No Change | 41
  Cycle 108: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 108: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 108: LVEF≥45% Points and Decr. from BL ≥10% Points | 8
  Cycle 111: number analyzed (Participants) | 42
  Cycle 111: Incr. or Decr. from BL <10% Points, or No Change | 34
  Cycle 111: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 111: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 111: LVEF≥45% Points and Decr. from BL ≥10% Points | 8
  Cycle 114: number analyzed (Participants) | 23
  Cycle 114: Incr. or Decr. from BL <10% Points, or No Change | 19
  Cycle 114: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 114: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 114: LVEF≥45% Points and Decr. from BL ≥10% Points | 4
  Cycle 117: number analyzed (Participants) | 17
  Cycle 117: Incr. or Decr. from BL <10% Points, or No Change | 11
  Cycle 117: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 117: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 117: LVEF≥45% Points and Decr. from BL ≥10% Points | 6
  Cycle 120: number analyzed (Participants) | 7
  Cycle 120: Incr. or Decr. from BL <10% Points, or No Change | 4
  Cycle 120: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 120: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 120: LVEF≥45% Points and Decr. from BL ≥10% Points | 3
  Cycle 123: number analyzed (Participants) | 3
  Cycle 123: Incr. or Decr. from BL <10% Points, or No Change | 2
  Cycle 123: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 123: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 123: LVEF≥45% Points and Decr. from BL ≥10% Points | 1
  Cycle 126: number analyzed (Participants) | 1
  Cycle 126: Incr. or Decr. from BL <10% Points, or No Change | 1
  Cycle 126: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 0
  Cycle 126: LVEF<45% Points and Decr. from BL ≥15% Points | 0
  Cycle 126: LVEF≥45% Points and Decr. from BL ≥10% Points | 0
  End of Treatment: number analyzed (Participants) | 546
  End of Treatment: Incr. or Decr. from BL <10% Points, or No Change | 431
  End of Treatment: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 2
  End of Treatment: LVEF<45% Points and Decr. from BL ≥15% Points | 26
  End of Treatment: LVEF≥45% Points and Decr. from BL ≥10% Points | 87
  Day 28 of Follow-Up: number analyzed (Participants) | 584
  Day 28 of Follow-Up: Incr. or Decr. from BL <10% Points, or No Change | 472
  Day 28 of Follow-Up: LVEF<45% Points and Decr. from BL ≥10%-<15% Points | 4
  Day 28 of Follow-Up: LVEF<45% Points and Decr. from BL ≥15% Points | 22
  Day 28 of Follow-Up: LVEF≥45% Points and Decr. from BL ≥10% Points | 86

24. Primary Outcome: Number of Participants With Laboratory Abnormalities in Hematology and Coagulation Parameters: Shift From Baseline to the Worst Post-Baseline Grade According to NCI-CTC v4.0
Description: Clinical laboratory tests for hematology and coagulation parameters were performed at local laboratories. Laboratory toxicities were defined based on NCI-CTC v4.0 from Grades 1 (least severe) to 4 (most severe). Some laboratory parameters are bi-dimensional (i.e. can be graded in both the low and high direction). These parameters were split and presented in both directions. Baseline was defined as the last non-missing measurement taken prior to the first dose of study treatment (including unscheduled assessments). Values from all visits, including unscheduled visits, were included in the derivation of the worst post-baseline grade. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: was clinically significant (per investigator); was accompanied by clinical symptoms; resulted in a change in study treatment; or resulted in a medical intervention or a change in concomitant therapy.
Time Frame: Predose at each treatment cycle (1 cycle is 3 weeks) from Baseline until 28 days after the last dose of study treatment. The median (full range) duration of exposure to any study treatment was 16.2 (0.0-86.4) months.
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Absolute Neutrophil Count: Normal to Normal | 844
  Absolute Neutrophil Count: Normal to Grade 1 | 232
  Absolute Neutrophil Count: Normal to Grade 2 | 169
  Absolute Neutrophil Count: Normal to Grade 3 | 45
  Absolute Neutrophil Count: Normal to Grade 4 | 27
  Absolute Neutrophil Count: Normal to Missing | 27
  Absolute Neutrophil Count: Grade 1 to Normal | 3
  Absolute Neutrophil Count: Grade 1 to 1 | 11
  Absolute Neutrophil Count: Grade 1 to 2 | 14
  Absolute Neutrophil Count: Grade 1 to 3 | 3
  Absolute Neutrophil Count: Grade 2 to 1 | 2
  Absolute Neutrophil Count: Missing to Normal | 21
  Absolute Neutrophil Count: Missing to Grade 1 | 2
  Absolute Neutrophil Count: Missing to Grade 2 | 3
  Absolute Neutrophil Count: Missing to Grade 4 | 1
  Absolute Neutrophil Count: Missing to Missing | 32
  Hemoglobin (High): Normal to Normal | 1327
  Hemoglobin (High): Normal to Grade 1 | 29
  Hemoglobin (High): Normal to Grade 3 | 1
  Hemoglobin (High): Normal to Missing | 26
  Hemoglobin (High): Grade 1 to Normal | 28
  Hemoglobin (High): Grade 1 to 1 | 5
  Hemoglobin (High): Grade 1 to Missing | 2
  Hemoglobin (High): Grade 2 to Normal | 1
  Hemoglobin (High): Missing to Normal | 14
  Hemoglobin (High): Missing to Missing | 3
  Hemoglobin (Low): Normal to Normal | 257
  Hemoglobin (Low): Normal to Grade 1 | 648
  Hemoglobin (Low): Normal to Grade 2 | 198
  Hemoglobin (Low): Normal to Grade 3 | 10
  Hemoglobin (Low): Normal to Missing | 21
  Hemoglobin (Low): Grade 1 to Normal | 2
  Hemoglobin (Low): Grade 1 to 1 | 109
  Hemoglobin (Low): Grade 1 to 2 | 128
  Hemoglobin (Low): Grade 1 to 3 | 12
  Hemoglobin (Low): Grade 1 to Missing | 4
  Hemoglobin (Low): Grade 2 to 1 | 5
  Hemoglobin (Low): Grade 2 to 2 | 18
  Hemoglobin (Low): Grade 2 to 3 | 3
  Hemoglobin (Low): Grade 2 to Missing | 3
  Hemoglobin (Low): Grade 3 to 1 | 1
  Hemoglobin (Low): Missing to Normal | 3
  Hemoglobin (Low): Missing to Grade 1 | 7
  Hemoglobin (Low): Missing to Grade 2 | 4
  Hemoglobin (Low): Missing to Missing | 3
  Lymphocytes (High): Normal to Normal | 1251
  Lymphocytes (High): Normal to Grade 2 | 111
  Lymphocytes (High): Normal to Grade 3 | 8
  Lymphocytes (High): Normal to Missing | 28
  Lymphocytes (High): Grade 2 to Normal | 4
  Lymphocytes (High): Grade 2 to 2 | 10
  Lymphocytes (High): Grade 2 to 3 | 2
  Lymphocytes (High): Grade 3 to Normal | 1
  Lymphocytes (High): Grade 3 to 3 | 2
  Lymphocytes (High): Missing to Normal | 15
  Lymphocytes (High): Missing to Grade 2 | 2
  Lymphocytes (High): Missing to Missing | 2
  Lymphocytes (Low): Normal to Normal | 565
  Lymphocytes (Low): Normal to Grade 1 | 255
  Lymphocytes (Low): Normal to Grade 2 | 210
  Lymphocytes (Low): Normal to Grade 3 | 76
  Lymphocytes (Low): Normal to Grade 4 | 18
  Lymphocytes (Low): Normal to Missing | 19
  Lymphocytes (Low): Grade 1 to Normal | 11
  Lymphocytes (Low): Grade 1 to 1 | 54
  Lymphocytes (Low): Grade 1 to 2 | 51
  Lymphocytes (Low): Grade 1 to 3 | 18
  Lymphocytes (Low): Grade 1 to 4 | 6
  Lymphocytes (Low): Grade 1 to Missing | 5
  Lymphocytes (Low): Grade 2 to Normal | 12
  Lymphocytes (Low): Grade 2 to 1 | 8
  Lymphocytes (Low): Grade 2 to 2 | 37
  Lymphocytes (Low): Grade 2 to 3 | 19
  Lymphocytes (Low): Grade 2 to 4 | 1
  Lymphocytes (Low): Grade 2 to Missing | 2
  Lymphocytes (Low): Grade 3 to 1 | 3
  Lymphocytes (Low): Grade 3 to 2 | 8
  Lymphocytes (Low): Grade 3 to 3 | 14
  Lymphocytes (Low): Grade 3 to 4 | 2
  Lymphocytes (Low): Grade 3 to Missing | 1
  Lymphocytes (Low): Grade 4 to 2 | 1
  Lymphocytes (Low): Grade 4 to 3 | 3
  Lymphocytes (Low): Grade 4 to 4 | 16
  Lymphocytes (Low): Grade 4 to Missing | 1
  Lymphocytes (Low): Missing to Normal | 11
  Lymphocytes (Low): Missing to Grade 1 | 3
  Lymphocytes (Low): Missing to Grade 2 | 3
  Lymphocytes (Low): Missing to Grade 3 | 1
  Lymphocytes (Low): Missing to Missing | 2
  Platelet Count: Normal to Normal | 1222
  Platelet Count: Normal to Grade 1 | 149
  Platelet Count: Normal to Grade 3 | 1
  Platelet Count: Normal to Grade 4 | 2
  Platelet Count: Normal to Missing | 26
  Platelet Count: Grade 1 to Normal | 15
  Platelet Count: Grade 1 to 1 | 16
  Platelet Count: Grade 1 to 2 | 1
  Platelet Count: Grade 1 to Missing | 2
  Platelet Count: Missing to Normal | 1
  Platelet Count: Missing to Grade 1 | 1
  White Blood Cells (High): Normal to Normal | 1391
  White Blood Cells (High): Normal to Missing | 29
  White Blood Cells (High): Missing to Normal | 14
  White Blood Cells (High): Missing to Missing | 2
  White Blood Cells (Low): Normal to Normal | 702
  White Blood Cells (Low): Normal to Grade 1 | 392
  White Blood Cells (Low): Normal to Grade 2 | 190
  White Blood Cells (Low): Normal to Grade 3 | 29
  White Blood Cells (Low): Normal to Grade 4 | 6
  White Blood Cells (Low): Normal to Missing | 29
  White Blood Cells (Low): Grade 1 to Normal | 4
  White Blood Cells (Low): Grade 1 to 1 | 20
  White Blood Cells (Low): Grade 1 to 2 | 33
  White Blood Cells (Low): Grade 1 to 3 | 4
  White Blood Cells (Low): Grade 2 to Normal | 2
  White Blood Cells (Low): Grade 2 to 1 | 4
  White Blood Cells (Low): Grade 2 to 2 | 3
  White Blood Cells (Low): Grade 3 to Normal | 1
  White Blood Cells (Low): Grade 3 to 3 | 1
  White Blood Cells (Low): Missing to Normal | 9
  White Blood Cells (Low): Missing to Grade 1 | 3
  White Blood Cells (Low): Missing to Grade 2 | 1
  White Blood Cells (Low): Missing to Grade 3 | 1
  White Blood Cells (Low): Missing to Missing | 2
  International Normalized Ratio: Normal to Normal | 17
  International Normalized Ratio: Normal to Grade 1 | 52
  International Normalized Ratio: Normal to Grade 2 | 1
  International Normalized Ratio: Normal to Missing | 3
  International Normalized Ratio: Grade 1 to Normal | 1
  International Normalized Ratio: Grade 2 to 3 | 1
  International Normalized Ratio: Missing to Normal | 424
  International Normalized Ratio: Missing to Grade 1 | 615
  International Normalized Ratio: Missing to Grade 2 | 23
  International Normalized Ratio: Missing to Grade 3 | 14
  International Normalized Ratio: Missing to Missing | 285

25. Primary Outcome: Number of Participants With Laboratory Abnormalities in Hematology and Coagulation Parameters: Shift From Baseline to the Worst Post-Baseline Grade According to Normal Range Criteria
Description: Clinical laboratory tests for hematology and coagulation parameters were performed at local laboratories. Laboratory toxicities were defined based on local laboratory normal ranges (for parameters with NCI-CTC grade not defined). Some laboratory parameters are bi-dimensional (i.e. can be graded in both the low and high direction). These parameters were split and presented in both directions. Baseline was defined as the last non-missing measurement taken prior to the first dose of study treatment (including unscheduled assessments). Values from all visits, including unscheduled visits, were included in the derivation of the worst post-baseline grade. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: was clinically significant (per investigator); was accompanied by clinical symptoms; resulted in a change in study treatment; or resulted in a medical intervention or a change in concomitant therapy.
Time Frame: as for outcome 24
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Basophils (High): Normal to Normal | 1020
  Basophils (High): Normal to Low | 3
  Basophils (High): Normal to High | 261
  Basophils (High): Low to Normal | 16
  Basophils (High): Low to Low | 1
  Basophils (High): Low to High | 5
  Basophils (High): High to Normal | 11
  Basophils (High): High to High | 38
  Basophils (High): Missing to Normal | 21
  Basophils (High): Missing to High | 7
  Basophils (High): Missing to Missing | 53
  Basophils (Low): Normal to Normal | 1206
  Basophils (Low): Normal to Low | 77
  Basophils (Low): Normal to High | 1
  Basophils (Low): Low to Normal | 3
  Basophils (Low): Low to Low | 18
  Basophils (Low): Low to Missing | 1
  Basophils (Low): High to Normal | 36
  Basophils (Low): High to Low | 5
  Basophils (Low): High to High | 8
  Basophils (Low): Missing to Normal | 40
  Basophils (Low): Missing to Low | 3
  Basophils (Low): Missing to High | 1
  Basophils (Low): Missing to Missing | 37
  Eosinophils (High): Normal to Normal | 904
  Eosinophils (High): Normal to Low | 13
  Eosinophils (High): Normal to High | 283
  Eosinophils (High): Low to Normal | 66
  Eosinophils (High): Low to Low | 13
  Eosinophils (High): Low to High | 36
  Eosinophils (High): High to Normal | 11
  Eosinophils (High): High to High | 35
  Eosinophils (High): Missing to Normal | 17
  Eosinophils (High): Missing to Low | 1
  Eosinophils (High): Missing to High | 7
  Eosinophils (High): Missing to Missing | 50
  Eosinophils (Low): Normal to Normal | 810
  Eosinophils (Low): Normal to Low | 390
  Eosinophils (Low): Low to Normal | 13
  Eosinophils (Low): Low to Low | 101
  Eosinophils (Low): Low to High | 1
  Eosinophils (Low): High to Normal | 28
  Eosinophils (Low): High to Low | 13
  Eosinophils (Low): High to High | 5
  Eosinophils (Low): Missing to Normal | 37
  Eosinophils (Low): Missing to Low | 10
  Eosinophils (Low): Missing to Missing | 28
  Hematocrit (High): Normal to Normal | 953
  Hematocrit (High): Normal to Low | 47
  Hematocrit (High): Normal to High | 58
  Hematocrit (High): Normal to Missing | 4
  Hematocrit (High): Low to Normal | 201
  Hematocrit (High): Low to Low | 97
  Hematocrit (High): Low to High | 10
  Hematocrit (High): Low to Missing | 2
  Hematocrit (High): High to Normal | 17
  Hematocrit (High): High to High | 12
  Hematocrit (High): Missing to Normal | 15
  Hematocrit (High): Missing to High | 1
  Hematocrit (High): Missing to Missing | 19
  Hematocrit (Low): Normal to Normal | 223
  Hematocrit (Low): Normal to Low | 837
  Hematocrit (Low): Normal to Missing | 2
  Hematocrit (Low): Low to Normal | 5
  Hematocrit (Low): Low to Low | 305
  Hematocrit (Low): High to Normal | 13
  Hematocrit (Low): High to Low | 16
  Hematocrit (Low): Missing to Normal | 3
  Hematocrit (Low): Missing to Low | 12
  Hematocrit (Low): Missing to Missing | 20
  Monocytes (High): Normal to Normal | 802
  Monocytes (High): Normal to Low | 3
  Monocytes (High): Normal to High | 365
  Monocytes (High): Low to Normal | 58
  Monocytes (High): Low to Low | 6
  Monocytes (High): Low to High | 17
  Monocytes (High): High to Normal | 29
  Monocytes (High): High to Low | 1
  Monocytes (High): High to High | 82
  Monocytes (High): Missing to Normal | 12
  Monocytes (High): Missing to High | 8
  Monocytes (High): Missing to Missing | 53
  Monocytes (Low): Normal to Normal | 747
  Monocytes (Low): Normal to Low | 420
  Monocytes (Low): Normal to High | 3
  Monocytes (Low): Low to Normal | 11
  Monocytes (Low): Low to Low | 70
  Monocytes (Low): High to Normal | 64
  Monocytes (Low): High to Low | 40
  Monocytes (Low): High to High | 8
  Monocytes (Low): Missing to Normal | 13
  Monocytes (Low): Missing to Low | 10
  Monocytes (Low): Missing to High | 5
  Monocytes (Low): Missing to Missing | 45
  Red Blood Cells (High): Normal to Normal | 975
  Red Blood Cells (High): Normal to Low | 31
  Red Blood Cells (High): Normal to High | 111
  Red Blood Cells (High): Low to Normal | 131
  Red Blood Cells (High): Low to Low | 61
  Red Blood Cells (High): Low to High | 15
  Red Blood Cells (High): High to Normal | 22
  Red Blood Cells (High): High to High | 45
  Red Blood Cells (High): Missing to Normal | 18
  Red Blood Cells (High): Missing to Low | 2
  Red Blood Cells (High): Missing to High | 2
  Red Blood Cells (High): Missing to Missing | 23
  Red Blood Cells (Low): Normal to Normal | 350
  Red Blood Cells (Low): Normal to Low | 767
  Red Blood Cells (Low): Low to Normal | 10
  Red Blood Cells (Low): Low to Low | 197
  Red Blood Cells (Low): High to Normal | 44
  Red Blood Cells (Low): High to Low | 21
  Red Blood Cells (Low): High to High | 2
  Red Blood Cells (Low): Missing to Normal | 6
  Red Blood Cells (Low): Missing to Low | 16
  Red Blood Cells (Low): Missing to Missing | 23
  PTT (High): Normal to Normal | 46
  PTT (High): Normal to Low | 1
  PTT (High): Normal to High | 15
  PTT (High): Low to Normal | 19
  PTT (High): Low to Low | 1
  PTT (High): Low to High | 1
  PTT (High): High to High | 1
  PTT (High): Missing to Normal | 19
  PTT (High): Missing to Low | 5
  PTT (High): Missing to High | 9
  PTT (High): Missing to Missing | 1319
  PTT (Low): Normal to Normal | 46
  PTT (Low): Normal to Low | 16
  PTT (Low): Low to Normal | 3
  PTT (Low): Low to Low | 18
  PTT (Low): High to Normal | 1
  PTT (Low): Missing to Normal | 20
  PTT (Low): Missing to Low | 6
  PTT (Low): Missing to High | 5
  PTT (Low): Missing to Missing | 1321

26. Primary Outcome: Number of Participants With Laboratory Abnormalities in Biochemistry Parameters: Shift From Baseline to the Worst Post-Baseline Grade According to NCI-CTC v4.0
Description: Clinical laboratory tests for biochemistry parameters were performed at local laboratories. Laboratory toxicities were defined based on NCI-CTC v4.0 from Grades 1 (least severe) to 4 (most severe). Some laboratory parameters are bi-dimensional (i.e. can be graded in both the low and high direction). These parameters were split and presented in both directions. Baseline was defined as the last non-missing measurement taken prior to the first dose of study treatment (including unscheduled assessments). Values from all visits, including unscheduled visits, were included in the derivation of the worst post-baseline grade. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: was clinically significant (per investigator); was accompanied by clinical symptoms; resulted in a change in study treatment; or resulted in a medical intervention or a change in concomitant therapy.
Time Frame: as for outcome 24
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Alanine Aminotransferase: Normal to Normal | 610
  Alanine Aminotransferase: Normal to Grade 1 | 425
  Alanine Aminotransferase: Normal to Grade 2 | 26
  Alanine Aminotransferase: Normal to Grade 3 | 19
  Alanine Aminotransferase: Normal to Missing | 25
  Alanine Aminotransferase: Grade 1 to Normal | 75
  Alanine Aminotransferase: Grade 1 to 1 | 151
  Alanine Aminotransferase: Grade 1 to 2 | 26
  Alanine Aminotransferase: Grade 1 to 3 | 14
  Alanine Aminotransferase: Grade 1 to Missing | 6
  Alanine Aminotransferase: Grade 2 to Normal | 8
  Alanine Aminotransferase: Grade 2 to 1 | 28
  Alanine Aminotransferase: Grade 2 to 2 | 5
  Alanine Aminotransferase: Grade 2 to 3 | 1
  Alanine Aminotransferase: Grade 3 to 1 | 2
  Alanine Aminotransferase: Missing to Normal | 7
  Alanine Aminotransferase: Missing to Grade 1 | 4
  Alanine Aminotransferase: Missing to Grade 2 | 1
  Alanine Aminotransferase: Missing to Missing | 3
  Aspartate Aminotransferase: Normal to Normal | 562
  Aspartate Aminotransferase: Normal to Grade 1 | 386
  Aspartate Aminotransferase: Normal to Grade 2 | 22
  Aspartate Aminotransferase: Normal to Grade 3 | 9
  Aspartate Aminotransferase: Normal to Missing | 15
  Aspartate Aminotransferase: Grade 1 to Normal | 120
  Aspartate Aminotransferase: Grade 1 to 1 | 187
  Aspartate Aminotransferase: Grade 1 to 2 | 24
  Aspartate Aminotransferase: Grade 1 to 3 | 9
  Aspartate Aminotransferase: Grade 1 to Missing | 14
  Aspartate Aminotransferase: Grade 2 to Normal | 13
  Aspartate Aminotransferase: Grade 2 to 1 | 29
  Aspartate Aminotransferase: Grade 2 to 2 | 3
  Aspartate Aminotransferase: Grade 2 to Missing | 3
  Aspartate Aminotransferase: Grade 3 to Normal | 2
  Aspartate Aminotransferase: Grade 3 to 1 | 7
  Aspartate Aminotransferase: Grade 3 to Missing | 1
  Aspartate Aminotransferase: Missing to Normal | 13
  Aspartate Aminotransferase: Missing to Grade 1 | 9
  Aspartate Aminotransferase: Missing to Grade 2 | 2
  Aspartate Aminotransferase: Missing to Missing | 6
  Albumin: Normal to Normal | 785
  Albumin: Normal to Grade 1 | 357
  Albumin: Normal to Grade 2 | 86
  Albumin: Normal to Grade 3 | 10
  Albumin: Normal to Missing | 23
  Albumin: Grade 1 to Normal | 13
  Albumin: Grade 1 to 1 | 43
  Albumin: Grade 1 to 2 | 35
  Albumin: Grade 1 to 3 | 1
  Albumin: Grade 1 to Missing | 7
  Albumin: Grade 2 to Normal | 3
  Albumin: Grade 2 to 1 | 5
  Albumin: Grade 2 to 2 | 8
  Albumin: Grade 2 to 3 | 2
  Albumin: Grade 2 to Missing | 2
  Albumin: Grade 3 to 2 | 1
  Albumin: Grade 3 to Missing | 1
  Albumin: Missing to Normal | 28
  Albumin: Missing to Grade 1 | 14
  Albumin: Missing to Grade 2 | 6
  Albumin: Missing to Missing | 6
  Alkaline Phosphatase: Normal to Normal | 605
  Alkaline Phosphatase: Normal to Grade 1 | 329
  Alkaline Phosphatase: Normal to Grade 2 | 14
  Alkaline Phosphatase: Normal to Grade 3 | 2
  Alkaline Phosphatase: Normal to Missing | 18
  Alkaline Phosphatase: Grade 1 to Normal | 44
  Alkaline Phosphatase: Grade 1 to 1 | 241
  Alkaline Phosphatase: Grade 1 to 2 | 72
  Alkaline Phosphatase: Grade 1 to 3 | 15
  Alkaline Phosphatase: Grade 1 to Missing | 6
  Alkaline Phosphatase: Grade 2 to Normal | 2
  Alkaline Phosphatase: Grade 2 to 1 | 21
  Alkaline Phosphatase: Grade 2 to 2 | 24
  Alkaline Phosphatase: Grade 2 to 3 | 14
  Alkaline Phosphatase: Grade 2 to Missing | 8
  Alkaline Phosphatase: Grade 3 to 1 | 2
  Alkaline Phosphatase: Grade 3 to 2 | 1
  Alkaline Phosphatase: Grade 3 to 3 | 4
  Alkaline Phosphatase: Missing to Normal | 7
  Alkaline Phosphatase: Missing to Grade 1 | 3
  Alkaline Phosphatase: Missing to Grade 3 | 1
  Alkaline Phosphatase: Missing to Missing | 3
  Calcium (High): Normal to Normal | 1060
  Calcium (High): Normal to Grade 1 | 192
  Calcium (High): Normal to Grade 2 | 2
  Calcium (High): Normal to Grade 3 | 1
  Calcium (High): Normal to Grade 4 | 1
  Calcium (High): Normal to Missing | 26
  Calcium (High): Grade 1 to Normal | 47
  Calcium (High): Grade 1 to 1 | 47
  Calcium (High): Grade 1 to 2 | 1
  Calcium (High): Grade 1 to 3 | 1
  Calcium (High): Grade 1 to Missing | 5
  Calcium (High): Grade 2 to Normal | 1
  Calcium (High): Grade 2 to 1 | 1
  Calcium (High): Grade 2 to 2 | 1
  Calcium (High): Grade 3 to Normal | 2
  Calcium (High): Grade 3 to 1 | 1
  Calcium (High): Grade 3 to 2 | 1
  Calcium (High): Grade 4 to Normal | 1
  Calcium (High): Missing to Normal | 32
  Calcium (High): Missing to Grade 1 | 3
  Calcium (High): Missing to Missing | 10
  Calcium (Low): Normal to Normal | 786
  Calcium (Low): Normal to Grade 1 | 378
  Calcium (Low): Normal to Grade 2 | 117
  Calcium (Low): Normal to Grade 3 | 18
  Calcium (Low): Normal to Missing | 30
  Calcium (Low): Grade 1 to Normal | 5
  Calcium (Low): Grade 1 to 1 | 31
  Calcium (Low): Grade 1 to 2 | 12
  Calcium (Low): Grade 1 to 3 | 2
  Calcium (Low): Grade 1 to Missing | 1
  Calcium (Low): Grade 2 to Normal | 5
  Calcium (Low): Grade 2 to 1 | 1
  Calcium (Low): Grade 2 to 2 | 4
  Calcium (Low): Grade 3 to 3 | 1
  Calcium (Low): Missing to Normal | 20
  Calcium (Low): Missing to Grade 1 | 11
  Calcium (Low): Missing to Grade 2 | 4
  Calcium (Low): Missing to Missing | 10
  Creatinine: Normal to Normal | 176
  Creatinine: Normal to Grade 1 | 960
  Creatinine: Normal to Grade 2 | 175
  Creatinine: Normal to Grade 3 | 5
  Creatinine: Normal to Grade 4 | 5
  Creatinine: Normal to Missing | 26
  Creatinine: Grade 1 to Normal | 12
  Creatinine: Grade 1 to 1 | 38
  Creatinine: Grade 1 to 2 | 8
  Creatinine: Grade 1 to Missing | 3
  Creatinine: Grade 2 to 2 | 3
  Creatinine: Grade 2 to 3 | 1
  Creatinine: Grade 2 to Missing | 1
  Creatinine: Missing to Normal | 11
  Creatinine: Missing to Grade 1 | 6
  Creatinine: Missing to Missing | 6
  Gamma-Glutamyl Transpeptidase: Normal to Normal | 498
  Gamma-Glutamyl Transpeptidase: Normal to Grade 1 | 227
  Gamma-Glutamyl Transpeptidase: Normal to Grade 2 | 39
  Gamma-Glutamyl Transpeptidase: Normal to Grade 3 | 15
  Gamma-Glutamyl Transpeptidase: Normal to Missing | 12
  Gamma-Glutamyl Transpeptidase: Grade 1 to Normal | 64
  Gamma-Glutamyl Transpeptidase: Grade 1 to 1 | 187
  Gamma-Glutamyl Transpeptidase: Grade 1 to 2 | 75
  Gamma-Glutamyl Transpeptidase: Grade 1 to 3 | 20
  Gamma-Glutamyl Transpeptidase: Grade 1 to Missing | 7
  Gamma-Glutamyl Transpeptidase: Grade 2 to Normal | 5
  Gamma-Glutamyl Transpeptidase: Grade 2 to 1 | 52
  Gamma-Glutamyl Transpeptidase: Grade 2 to 2 | 45
  Gamma-Glutamyl Transpeptidase: Grade 2 to 3 | 21
  Gamma-Glutamyl Transpeptidase: Grade 2 to Missing | 5
  Gamma-Glutamyl Transpeptidase: Grade 3 to Normal | 2
  Gamma-Glutamyl Transpeptidase: Grade 3 to 1 | 15
  Gamma-Glutamyl Transpeptidase: Grade 3 to 2 | 38
  Gamma-Glutamyl Transpeptidase: Grade 3 to 3 | 47
  Gamma-Glutamyl Transpeptidase: Grade 3 to Missing | 4
  Gamma-Glutamyl Transpeptidase: Missing to Normal | 14
  Gamma-Glutamyl Transpeptidase: Missing to Grade 1 | 7
  Gamma-Glutamyl Transpeptidase: Missing to Grade 2 | 10
  Gamma-Glutamyl Transpeptidase: Missing to Grade 3 | 18
  Gamma-Glutamyl Transpeptidase: Missing to Missing | 9
  Glucose (High): Normal to Normal | 340
  Glucose (High): Normal to Grade 1 | 534
  Glucose (High): Normal to Grade 2 | 115
  Glucose (High): Normal to Missing | 21
  Glucose (High): Grade 1 to Normal | 28
  Glucose (High): Grade 1 to 1 | 190
  Glucose (High): Grade 1 to 2 | 74
  Glucose (High): Grade 1 to Missing | 9
  Glucose (High): Grade 2 to Normal | 2
  Glucose (High): Grade 2 to 1 | 13
  Glucose (High): Grade 2 to 2 | 10
  Glucose (High): Grade 2 to Missing | 3
  Glucose (High): Missing to Normal | 20
  Glucose (High): Missing to Grade 1 | 30
  Glucose (High): Missing to Grade 2 | 40
  Glucose (High): Missing to Missing | 7
  Glucose (Low): Normal to Normal | 1061
  Glucose (Low): Normal to Grade 1 | 173
  Glucose (Low): Normal to Grade 2 | 19
  Glucose (Low): Normal to Grade 3 | 4
  Glucose (Low): Normal to Grade 4 | 5
  Glucose (Low): Normal to Missing | 33
  Glucose (Low): Grade 1 to Normal | 8
  Glucose (Low): Grade 1 to 1 | 24
  Glucose (Low): Grade 1 to 2 | 3
  Glucose (Low): Grade 1 to 3 | 1
  Glucose (Low): Grade 1 to 4 | 1
  Glucose (Low): Grade 2 to Normal | 1
  Glucose (Low): Missing to Normal | 69
  Glucose (Low): Missing to Grade 1 | 16
  Glucose (Low): Missing to Grade 2 | 2
  Glucose (Low): Missing to Grade 3 | 1
  Glucose (Low): Missing to Missing | 15
  Magnesium (High): Normal to Normal | 1100
  Magnesium (High): Normal to Grade 1 | 122
  Magnesium (High): Normal to Grade 3 | 38
  Magnesium (High): Normal to Grade 4 | 6
  Magnesium (High): Normal to Missing | 31
  Magnesium (High): Grade 1 to Normal | 12
  Magnesium (High): Grade 1 to 1 | 7
  Magnesium (High): Grade 3 to Normal | 2
  Magnesium (High): Grade 3 to 3 | 2
  Magnesium (High): Grade 4 to Normal | 1
  Magnesium (High): Grade 4 to 4 | 1
  Magnesium (High): Missing to Normal | 85
  Magnesium (High): Missing to Grade 1 | 12
  Magnesium (High): Missing to Grade 3 | 6
  Magnesium (High): Missing to Missing | 11
  Magnesium (Low): Normal to Normal | 857
  Magnesium (Low): Normal to Grade 1 | 319
  Magnesium (Low): Normal to Grade 2 | 28
  Magnesium (Low): Normal to Grade 3 | 9
  Magnesium (Low): Normal to Grade 4 | 3
  Magnesium (Low): Normal to Missing | 28
  Magnesium (Low): Grade 1 to Normal | 9
  Magnesium (Low): Grade 1 to 1 | 55
  Magnesium (Low): Grade 1 to 2 | 7
  Magnesium (Low): Grade 1 to 3 | 3
  Magnesium (Low): Grade 1 to Missing | 3
  Magnesium (Low): Grade 4 to 4 | 1
  Magnesium (Low): Missing to Normal | 81
  Magnesium (Low): Missing to Grade 1 | 19
  Magnesium (Low): Missing to Grade 2 | 1
  Magnesium (Low): Missing to Grade 3 | 1
  Magnesium (Low): Missing to Grade 4 | 1
  Magnesium (Low): Missing to Missing | 11
  Potassium (High): Normal to Normal | 1051
  Potassium (High): Normal to Grade 1 | 183
  Potassium (High): Normal to Grade 2 | 81
  Potassium (High): Normal to Grade 3 | 18
  Potassium (High): Normal to Grade 4 | 8
  Potassium (High): Normal to Missing | 26
  Potassium (High): Grade 1 to Normal | 16
  Potassium (High): Grade 1 to 1 | 8
  Potassium (High): Grade 1 to 2 | 7
  Potassium (High): Grade 1 to 3 | 1
  Potassium (High): Grade 1 to Missing | 3
  Potassium (High): Grade 2 to Normal | 2
  Potassium (High): Grade 2 to 1 | 1
  Potassium (High): Grade 2 to 2 | 1
  Potassium (High): Grade 4 to Normal | 1
  Potassium (High): Missing to Normal | 18
  Potassium (High): Missing to Grade 1 | 5
  Potassium (High): Missing to Grade 2 | 3
  Potassium (High): Missing to Missing | 3
  Potassium (Low): Normal to Normal | 990
  Potassium (Low): Normal to Grade 2 | 367
  Potassium (Low): Normal to Missing | 29
  Potassium (Low): Grade 2 to Normal | 8
  Potassium (Low): Grade 2 to 2 | 13
  Potassium (Low): Missing to Normal | 19
  Potassium (Low): Missing to Grade 2 | 7
  Potassium (Low): Missing to Missing | 3
  Sodium (High): Normal to Normal | 1075
  Sodium (High): Normal to Grade 1 | 256
  Sodium (High): Normal to Grade 2 | 36
  Sodium (High): Normal to Grade 3 | 9
  Sodium (High): Normal to Grade 4 | 1
  Sodium (High): Normal to Missing | 28
  Sodium (High): Grade 1 to Normal | 3
  Sodium (High): Grade 1 to 1 | 6
  Sodium (High): Grade 1 to 2 | 3
  Sodium (High): Grade 1 to 3 | 1
  Sodium (High): Grade 2 to 2 | 2
  Sodium (High): Grade 2 to 3 | 1
  Sodium (High): Grade 3 to Normal | 1
  Sodium (High): Grade 3 to Missing | 1
  Sodium (High): Missing to Normal | 11
  Sodium (High): Missing to Grade 1 | 1
  Sodium (High): Missing to Missing | 1
  Sodium (Low): Normal to Normal | 994
  Sodium (Low): Normal to Grade 1 | 298
  Sodium (Low): Normal to Grade 3 | 20
  Sodium (Low): Normal to Grade 4 | 15
  Sodium (Low): Normal to Missing | 23
  Sodium (Low): Grade 1 to Normal | 21
  Sodium (Low): Grade 1 to 1 | 36
  Sodium (Low): Grade 1 to 3 | 2
  Sodium (Low): Grade 1 to 4 | 1
  Sodium (Low): Grade 1 to Missing | 6
  Sodium (Low): Grade 3 to Normal | 1
  Sodium (Low): Grade 3 to 1 | 2
  Sodium (Low): Grade 3 to 3 | 1
  Sodium (Low): Grade 4 to Normal | 2
  Sodium (Low): Grade 4 to 1 | 1
  Sodium (Low): Missing to Normal | 6
  Sodium (Low): Missing to Grade 1 | 5
  Sodium (Low): Missing to Grade 3 | 1
  Sodium (Low): Missing to Missing | 1
  Total Bilirubin: Normal to Normal | 1231
  Total Bilirubin: Normal to Grade 1 | 88
  Total Bilirubin: Normal to Grade 2 | 35
  Total Bilirubin: Normal to Grade 3 | 2
  Total Bilirubin: Normal to Missing | 28
  Total Bilirubin: Grade 1 to Normal | 3
  Total Bilirubin: Grade 1 to 1 | 11
  Total Bilirubin: Grade 1 to 2 | 6
  Total Bilirubin: Grade 1 to Missing | 2
  Total Bilirubin: Grade 2 to 1 | 1
  Total Bilirubin: Grade 2 to 2 | 1
  Total Bilirubin: Grade 2 to Missing | 1
  Total Bilirubin: Grade 3 to Normal | 1
  Total Bilirubin: Missing to Normal | 22
  Total Bilirubin: Missing to Grade 2 | 1
  Total Bilirubin: Missing to Missing | 3
  Uric Acid: Normal to Normal | 933
  Uric Acid: Normal to Grade 1 | 190
  Uric Acid: Normal to Grade 4 | 8
  Uric Acid: Normal to Missing | 20
  Uric Acid: Grade 1 to Normal | 58
  Uric Acid: Grade 1 to 1 | 120
  Uric Acid: Grade 1 to 4 | 6
  Uric Acid: Grade 1 to Missing | 11
  Uric Acid: Grade 4 to Normal | 1
  Uric Acid: Grade 4 to 1 | 2
  Uric Acid: Grade 4 to 4 | 4
  Uric Acid: Grade 4 to Missing | 1
  Uric Acid: Missing to Normal | 57
  Uric Acid: Missing to Grade 1 | 13
  Uric Acid: Missing to Grade 4 | 2
  Uric Acid: Missing to Missing | 10

27. Primary Outcome: Number of Participants With Laboratory Abnormalities in Biochemistry Parameters: Shift From Baseline to the Worst Post-Baseline Grade According to Normal Range Criteria
Description: Clinical laboratory tests for biochemistry parameters were performed at local laboratories. Laboratory toxicities were defined based on local laboratory normal ranges (for parameters with NCI-CTC grade not defined). Some laboratory parameters are bi-dimensional (i.e. can be graded in both the low and high direction). These parameters were split and presented in both directions. Baseline was defined as the last non-missing measurement taken prior to the first dose of study treatment (including unscheduled assessments). Values from all visits, including unscheduled visits, were included in the derivation of the worst post-baseline grade. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: was clinically significant (per investigator); was accompanied by clinical symptoms; resulted in a change in study treatment; or resulted in a medical intervention or a change in concomitant therapy.
Time Frame: as for outcome 24
Population: Safety Population: all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Participants
  Blood Urea Nitrogen (High): Normal to Normal | 717
  Blood Urea Nitrogen (High): Normal to Low | 5
  Blood Urea Nitrogen (High): Normal to High | 402
  Blood Urea Nitrogen (High): Normal to Missing | 2
  Blood Urea Nitrogen (High): Low to Normal | 69
  Blood Urea Nitrogen (High): Low to Low | 8
  Blood Urea Nitrogen (High): Low to High | 12
  Blood Urea Nitrogen (High): High to Normal | 23
  Blood Urea Nitrogen (High): High to High | 98
  Blood Urea Nitrogen (High): Missing to Normal | 42
  Blood Urea Nitrogen (High): Missing to High | 19
  Blood Urea Nitrogen (High): Missing to Missing | 39
  Blood Urea Nitrogen (Low): Normal to Normal | 828
  Blood Urea Nitrogen (Low): Normal to Low | 293
  Blood Urea Nitrogen (Low): Normal to High | 3
  Blood Urea Nitrogen (Low): Normal to Missing | 2
  Blood Urea Nitrogen (Low): Low to Normal | 17
  Blood Urea Nitrogen (Low): Low to Low | 72
  Blood Urea Nitrogen (Low): High to Normal | 104
  Blood Urea Nitrogen (Low): High to Low | 11
  Blood Urea Nitrogen (Low): High to High | 6
  Blood Urea Nitrogen (Low): Missing to Normal | 47
  Blood Urea Nitrogen (Low): Missing to Low | 11
  Blood Urea Nitrogen (Low): Missing to High | 3
  Blood Urea Nitrogen (Low): Missing to Missing | 39
  Calc Creatinine Clearance (High): Normal to Normal | 540
  Calc Creatinine Clearance (High): Normal to Low | 11
  Calc Creatinine Clearance (High): Normal to High | 201
  Calc Creatinine Clearance(High): Normal to Missing | 2
  Calc Creatinine Clearance (High): Low to Normal | 166
  Calc Creatinine Clearance (High): Low to Low | 107
  Calc Creatinine Clearance (High): Low to High | 34
  Calc Creatinine Clearance (High): Low to Missing | 1
  Calc Creatinine Clearance (High): High to Normal | 13
  Calc Creatinine Clearance (High): High to High | 101
  Calc Creatinine Clearance(High): Missing to Normal | 46
  Calc Creatinine Clearance (High): Missing to Low | 8
  Calc Creatinine Clearance (High): Missing to High | 11
  Calc Creatinine Clearance(High):Missing to Missing | 195
  Calc Creatinine Clearance (Low): Normal to Normal | 393
  Calc Creatinine Clearance (Low): Normal to Low | 353
  Calc Creatinine Clearance (Low): Normal to High | 8
  Calc Creatinine Clearance (Low): Low to Normal | 12
  Calc Creatinine Clearance (Low): Low to Low | 294
  Calc Creatinine Clearance (Low): Low to High | 1
  Calc Creatinine Clearance (Low): Low to Missing | 1
  Calc Creatinine Clearance (Low): High to Normal | 61
  Calc Creatinine Clearance (Low): High to Low | 36
  Calc Creatinine Clearance (Low): High to High | 17
  Calc Creatinine Clearance (Low): Missing to Normal | 66
  Calc Creatinine Clearance (Low): Missing to Low | 44
  Calc Creatinine Clearance (Low): Missing to High | 17
  Calc Creatinine Clearance(Low): Missing to Missing | 133
  Chloride (High): Normal to Normal | 665
  Chloride (High): Normal to Low | 2
  Chloride (High): Normal to High | 508
  Chloride (High): Low to Normal | 54
  Chloride (High): Low to High | 13
  Chloride (High): High to Normal | 4
  Chloride (High): High to High | 58
  Chloride (High): Missing to Normal | 41
  Chloride (High): Missing to High | 32
  Chloride (High): Missing to Missing | 59
  Chloride (Low): Normal to Normal | 971
  Chloride (Low): Normal to Low | 201
  Chloride (Low): Normal to High | 3
  Chloride (Low): Low to Normal | 31
  Chloride (Low): Low to Low | 36
  Chloride (Low): High to Normal | 57
  Chloride (Low): High to Low | 4
  Chloride (Low): High to High | 1
  Chloride (Low): Missing to Normal | 60
  Chloride (Low): Missing to Low | 13
  Chloride (Low): Missing to High | 1
  Chloride (Low): Missing to Missing | 58
  Lactate Dehydrogenase (High): Normal to Normal | 328
  Lactate Dehydrogenase (High): Normal to High | 499
  Lactate Dehydrogenase (High): Low to Normal | 10
  Lactate Dehydrogenase (High): Low to Low | 1
  Lactate Dehydrogenase (High): Low to High | 4
  Lactate Dehydrogenase (High): High to Normal | 74
  Lactate Dehydrogenase (High): High to High | 449
  Lactate Dehydrogenase (High): Missing to Normal | 16
  Lactate Dehydrogenase (High): Missing to High | 30
  Lactate Dehydrogenase (High): Missing to Missing | 25
  Lactate Dehydrogenase (Low): Normal to Normal | 716
  Lactate Dehydrogenase (Low): Normal to Low | 102
  Lactate Dehydrogenase (Low): Normal to High | 9
  Lactate Dehydrogenase (Low): Low to Normal | 5
  Lactate Dehydrogenase (Low): Low to Low | 9
  Lactate Dehydrogenase (Low): Low to High | 1
  Lactate Dehydrogenase (Low): High to Normal | 426
  Lactate Dehydrogenase (Low): High to Low | 31
  Lactate Dehydrogenase (Low): High to High | 66
  Lactate Dehydrogenase (Low): Missing to Normal | 39
  Lactate Dehydrogenase (Low): Missing to Low | 3
  Lactate Dehydrogenase (Low): Missing to High | 3
  Lactate Dehydrogenase (Low): Missing to Missing | 26
  Total Protein (High): Normal to Normal | 1091
  Total Protein (High): Normal to Low | 20
  Total Protein (High): Normal to High | 110
  Total Protein (High): Low to Normal | 72
  Total Protein (High): Low to Low | 14
  Total Protein (High): High to Normal | 28
  Total Protein (High): High to High | 24
  Total Protein (High): Missing to Normal | 38
  Total Protein (High): Missing to Low | 3
  Total Protein (High): Missing to High | 4
  Total Protein (High): Missing to Missing | 32
  Total Protein (Low): Normal to Normal | 530
  Total Protein (Low): Normal to Low | 691
  Total Protein (Low): Low to Normal | 4
  Total Protein (Low): Low to Low | 82
  Total Protein (Low): High to Normal | 41
  Total Protein (Low): High to Low | 11
  Total Protein (Low): Missing to Normal | 23
  Total Protein (Low): Missing to Low | 23
  Total Protein (Low): Missing to Missing | 31

28. Secondary Outcome: Progression-Free Survival, as Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Description: Progression-free survival (PFS) was defined as the time between the date of enrollment and the date of first radiographically documented progressive disease assessment (by the investigator using RECIST v1.1) or death, whichever occurred first. PFS was analyzed using a Kaplan-Meier approach. Participants who had neither progressed nor died at the time of clinical cut-off or who were lost to follow-up were censored at the date of the last evaluable tumor assessment (response assessment with the latest end date); if no post-baseline assessments were available, such participants were censored at Day 1. If a participant missed 2 or more consecutive visits, then they were censored at the last evaluable visit prior to the missed visits. Tumor assessments were performed every 3 cycles (1 cycle is 3 weeks) for up to 36 months and at least every 12 cycles thereafter during treatment, and at least every 36 weeks post-treatment (if progression-free after 36 months), until disease progression.
Time Frame: From date of enrollment until date of disease progression or death, whichever occurred first. The median (full range) duration of follow-up was 68.73 (0.03-87.29) months.
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Months | 20.67 [18.89 to 23.13]

29. Secondary Outcome: Subgroup Analysis by Region of Enrollment: Progression-Free Survival, as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 28
Time Frame: as for outcome 28
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Europe | Asia | North America | South America | Africa | Other (Australia)
Number analyzed (Participants) | 1009 | 177 | 34 | 121 | 71 | 24
Months | 19.38 [17.51 to 21.75] | 23.79 [15.90 to 28.85] | 25.17 [14.42 to 29.44] | 22.37 [17.51 to 32.72] | 22.83 [12.02 to 27.86] | NA [15.74 to NA] — The median and upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study.

30. Secondary Outcome: Subgroup Analysis by Age (≤65 vs. >65 Years): Progression-Free Survival, as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 28
Time Frame: as for outcome 28
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Age ≤65 Years | Age >65 Years
Number analyzed (Participants) | 1167 | 269
Months | 21.98 [19.65 to 24.25] | 14.72 [12.22 to 19.55]

31. Secondary Outcome: Subgroup Analysis by ECOG Performance Status at Baseline: Progression-Free Survival, as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 28
Time Frame: as for outcome 28
Population: ITT Population: all participants enrolled in the study. There were 2 participants with missing evaluations for ECOG performance status at baseline who were excluded from this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ECOG Performance Status 0 or 1 | ECOG Performance Status 2
Number analyzed (Participants) | 1371 | 63
Months | 21.49 [19.45 to 23.98] | 12.88 [8.67 to 15.90]

32. Secondary Outcome: Subgroup Analysis by Taxane Chemotherapy: Progression-Free Survival, as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 28
Time Frame: as for outcome 28
Population: ITT Population: all participants enrolled in the study. Only participants who received any taxane chemotherapy during the study were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Paclitaxel | Nab-Paclitaxel
Number analyzed (Participants) | 775 | 588 | 65
Months | 19.38 [16.92 to 22.11] | 23.23 [19.58 to 25.59] | 19.22 [11.70 to 37.09]

33. Secondary Outcome: Subgroup Analysis by Visceral Disease at Baseline: Progression-Free Survival, as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 28
Time Frame: as for outcome 28
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Visceral Disease | Non-Visceral Disease
Number analyzed (Participants) | 992 | 444
Months | 18.23 [16.13 to 20.57] | 27.24 [23.75 to 34.40]

34. Secondary Outcome: Subgroup Analysis by Prior (Neo)Adjuvant Chemotherapy: Progression-Free Survival, as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 28
Time Frame: as for outcome 28
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Prior (Neo)Adjuvant Chemotherapy | No Prior (Neo)Adjuvant Chemotherapy
Number analyzed (Participants) | 786 | 650
Months | 19.12 [16.59 to 21.49] | 23.49 [20.57 to 25.63]

35. Secondary Outcome: Subgroup Analysis by Hormone Receptor Status at Baseline: Progression-Free Survival, as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 28
Time Frame: as for outcome 28
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Hormone Receptor Positive | Hormone Receptor Negative | Hormone Receptor Status Unknown
Number analyzed (Participants) | 918 | 512 | 6
Months | 20.60 [18.53 to 23.82] | 20.73 [17.05 to 23.79] | 32.13 [11.63 to 61.57]

36. Secondary Outcome: Subgroup Analysis by Previous Trastuzumab Therapy: Progression-Free Survival, as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 28
Time Frame: as for outcome 28
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Previous Trastuzumab Therapy | No Previous Trastuzumab Therapy
Number analyzed (Participants) | 400 | 1036
Months | 15.38 [13.67 to 19.02] | 23.39 [20.67 to 25.00]

37. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from the date of enrollment until the date of death due to any cause. Overall survival was analyzed using a Kaplan-Meier approach. Participants who had not died were censored at the last date they were known to be alive. When it was not possible to confirm the full death date, partial death dates were imputed to: 01 June of that year if only the year was known, 15th of that month if only the month and year were known. If the imputed date was before the last known alive date, the last known alive date was used as the imputation.
Time Frame: From date of enrollment until death due to any cause. The median (full range) duration of follow-up was 68.73 (0.03-87.29) months.
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1436
Months | 65.31 [60.88 to 70.87]

38. Secondary Outcome: Subgroup Analysis by Region of Enrollment: Overall Survival
Description: as for outcome 37
Time Frame: as for outcome 37
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Europe | Asia | North America | South America | Africa | Other (Australia)
Number analyzed (Participants) | 1009 | 177 | 34 | 121 | 71 | 24
Months | 66.56 [61.90 to 73.49] | 63.57 [47.57 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study. | 55.56 [41.49 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study. | NA [49.84 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study. | 53.22 [33.35 to 63.87] | NA [44.16 to NA] — The median and upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study.

39. Secondary Outcome: Subgroup Analysis by Age (≤65 vs. >65 Years): Overall Survival
Description: as for outcome 37
Time Frame: as for outcome 37
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Age ≤65 Years | Age >65 Years
Number analyzed (Participants) | 1167 | 269
Months | 70.01 [64.33 to 81.08] | 50.10 [41.26 to 53.98]

40. Secondary Outcome: Subgroup Analysis by ECOG Performance Status at Baseline: Overall Survival
Description: as for outcome 37
Time Frame: as for outcome 37
Population: as for outcome 31
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ECOG Performance Status 0 or 1 | ECOG Performance Status 2
Number analyzed (Participants) | 1371 | 63
Months | 67.25 [63.44 to 76.52] | 31.15 [20.50 to 39.13]

41. Secondary Outcome: Subgroup Analysis by Taxane Chemotherapy: Overall Survival
Description: as for outcome 37
Time Frame: as for outcome 37
Population: as for outcome 32
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel | Paclitaxel | Nab-Paclitaxel
Number analyzed (Participants) | 775 | 588 | 65
Months | 66.53 [61.67 to 77.27] | 64.03 [56.61 to 72.25] | 70.87 [39.69 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study.

42. Secondary Outcome: Subgroup Analysis by Visceral Disease at Baseline: Overall Survival
Description: as for outcome 37
Time Frame: as for outcome 37
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Visceral Disease | Non-Visceral Disease
Number analyzed (Participants) | 992 | 444
Months | 57.10 [52.40 to 63.44] | 81.08 [71.66 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study.

43. Secondary Outcome: Subgroup Analysis by Prior (Neo)Adjuvant Chemotherapy: Overall Survival
Description: as for outcome 37
Time Frame: as for outcome 37
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Prior (Neo)Adjuvant Chemotherapy | No Prior (Neo)Adjuvant Chemotherapy
Number analyzed (Participants) | 786 | 650
Months | 57.10 [51.06 to 62.82] | 79.80 [71.79 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study.

44. Secondary Outcome: Subgroup Analysis by Hormone Receptor Status at Baseline: Overall Survival
Description: as for outcome 37
Time Frame: as for outcome 37
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Hormone Receptor Positive | Hormone Receptor Negative | Hormone Receptor Status Unknown
Number analyzed (Participants) | 918 | 512 | 6
Months | 66.66 [62.39 to 77.27] | 60.19 [52.34 to 67.71] | NA [16.13 to NA] — The median and upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study.

45. Secondary Outcome: Subgroup Analysis by Previous Trastuzumab Therapy: Overall Survival
Description: as for outcome 37
Time Frame: as for outcome 37
Population: ITT Population: all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Previous Trastuzumab Therapy | No Previous Trastuzumab Therapy
Number analyzed (Participants) | 400 | 1036
Months | 54.08 [48.66 to 60.75] | 73.50 [65.61 to NA] — The upper limit of the 95% confidence interval could not be calculated because not enough events had occurred during the study.

46. Secondary Outcome: Overall Response Rate (Complete Response or Partial Response) Based on Best Overall Response (Confirmed) as Assessed by the Investigator Using RECIST v1.1
Description: The overall response rate was defined as the percentage of participants with complete response (CR) or partial response (PR) as their best confirmed response (≥4 weeks later), as assessed by the investigator using RECIST v1.1 from the start of study treatment until disease progression/recurrence or death. Responses according to RECIST v1.1 are defined as follows: CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimetres (mm).; PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants without post-baseline tumor assessments were considered non-responders.
Time Frame: Assessed every 3 cycles (1 cycle is 3 weeks) up to 36 months, and at least every 12 cycles thereafter, until disease progression or death. The median (full range) duration of follow-up was 68.73 (0.03-87.29) months.
Population: Only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1198
Percentage of participants | 79.5 [77.07 to 81.72]

47. Secondary Outcome: Percentage of Participants by Best Overall Response as Assessed by the Investigator Using RECIST v1.1
Description: Best overall response (BOR) was defined as the best response recorded from the first dose of study treatment until disease progression/recurrence or death in the absence of disease progression. The hierarchy used to determine BOR: Complete Response (CR)>Partial Response (PR)>Stable Disease (SD)>Progressive Disease (PD)>Not Evaluable. Note that CR or PR was confirmed ≥4 weeks later. RECIST v1.1 responses are defined as follows: CR = Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 millimetres (mm).; PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum.; PD = At least 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study, and absolute increase of ≥5 mm.; SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 46
Population: Only participants with measurable disease at baseline were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1198
Percentage of participants
  Complete Response (Confirmed) | 14.6
  Partial Response (Confirmed) | 64.9
  Stable Disease | 15.3
  Progressive Disease | 4.2
  Not Evaluable | 1.1

48. Secondary Outcome: Subgroup Analysis by Age (≤65 vs. >65 Years): Overall Response Rate (Complete Response or Partial Response) Based on Best Overall Response (Confirmed) as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 46
Time Frame: as for outcome 46
Population: Only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Age ≤65 Years | Age >65 Years
Number analyzed (Participants) | 968 | 230
Percentage of participants | 81.7 [79.13 to 84.10] | 70.0 [63.63 to 75.85]

49. Secondary Outcome: Subgroup Analysis by Taxane Chemotherapy: Overall Response Rate (Complete Response or Partial Response) Based on Best Overall Response (Confirmed) as Assessed by the Investigator Using RECIST v1.1
Description: as for outcome 46
Time Frame: as for outcome 46
Population: Only participants with measurable disease at baseline and those who had received any taxane chemotherapy were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Docetaxel | Paclitaxel | Nab-Paclitaxel
Number analyzed (Participants) | 657 | 481 | 53
Percentage of participants | 78.4 [75.04 to 81.48] | 82.1 [78.40 to 85.44] | 77.4 [63.79 to 87.72]

50. Secondary Outcome: Clinical Benefit Rate (CR or PR, or SD for at Least 6 Months) Based on Best Overall Response as Assessed by the Investigator Using RECIST v.1.1
Description: The clinical benefit rate was defined as the percentage of participants whose best confirmed response (≥4 weeks later) was a complete response (CR) or partial response (PR), or stable disease (SD) that lasted at least 6 months, as assessed by the investigator using RECIST v1.1 from the start of study treatment until disease progression/recurrence or death. Clinical benefit responses according to RECIST v1.1 are defined as follows: CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimetres (mm).; PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.; SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least 20% increase in sum of diameters of target lesions and absolute increase of ≥5 mm), taking as reference the smallest sum diameters while on study.
Time Frame: Assessed every 3 cycles (1 cycle is 3 weeks) up to 36 months, and at least every 12 cycles thereafter, until disease progression. The median (full range) duration of follow-up was 68.73 (0.03-87.29) months.
Population: Only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1198
Percentage of participants | 86.2 [84.14 to 88.13]

51. Secondary Outcome: Duration of Response as Assessed by the Investigator Using RECIST v1.1
Description: Duration of response (DOR) was defined as the time from when a confirmed best overall response of complete response (CR) or partial response (PR) was first documented to first documented disease progression or death from any cause (whichever occurred first). DOR was analyzed using a Kaplan-Meier approach. Participants who had not progressed or died after having had a confirmed response were censored at the date of their last tumor measurement. Response was assessed every 3 cycles (1 cycle is 3 weeks) up to 36 months, and at least every 12 cycles thereafter until event occurrence or end of study. Responses according to RECIST v1.1 are defined as follows: CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimetres (mm).; PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first confirmed response (CR or PR) to first documented disease progression or death from any cause, whichever occurred first. The median (full range) duration of follow-up was 68.73 (0.03-87.29) months.
Population: Only participants with measurable disease at baseline and a documented confirmed response (CR or PR) were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 952
Months | 20.01 [18.20 to 22.21]

52. Secondary Outcome: Time to Response for Participants With Best Overall Response of Complete Response or Partial Response, as Assessed by the Investigator Using RECIST v1.1
Description: Time to response (TTR) was defined as the time from the first study treatment administration to the date of first confirmed response (CR or PR). TTR was analyzed using a Kaplan-Meier approach. Participants who did not have CR or PR were censored at the date of their last evaluable tumor assessment. Participants for whom no post-baseline tumor assessments were available were censored at Day 1. Responses according to RECIST v1.1 are defined as follows: CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimetres (mm).; PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first study treatment until date of first confirmed response (CR or PR). The median (full range) duration of follow-up was 68.73 (0.03-87.29) months.
Population: Only participants with measurable disease at baseline were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1198
Months | 2.464 [2.398 to 2.497]

53. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) Questionnaire Total Score Over the Course of the Study
Description: The FACT-B questionnaire (version 4) was administered only to female participants to assess quality of life in five subscales: physical, social, emotional, and functional well-being, and breast cancer. Participants were given a series of statements in each subscale and were asked to rate how true each statement was for them during the past 7 days on a 5-point scale ranging from 0 (not at all) to 4 (very much). The calculated FACT-B total score, ranging from 0 to 148, was the sum of the scores for each subscale, provided that at least 80% of the items had been answered; a higher score indicated a better quality of life. If any of the 5 subscale scores were missing, the total score was also set to missing. Baseline was defined as the last non-missing measurement taken prior to first dose of study treatment (including unscheduled assessments). Post-baseline values were summarized for planned visits only.
Time Frame: Baseline, every 3 cycles (1 cycle is 3 weeks) during treatment period, and 28 days post-treatment safety follow-up. The median (full range) duration of exposure to any study treatment was 16.2 (0.0-86.4) months.
Population: ITT Population: only enrolled female participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1429
Score on a scale
  Baseline (BL): Absolute Value at Visit: number analyzed (Participants) | 1306
  Baseline (BL): Absolute Value at Visit | 99.87 (20.548)
  Change from BL at Cycle 3: number analyzed (Participants) | 1158
  Change from BL at Cycle 3 | 0.40 (15.526)
  Change from BL at Cycle 6: number analyzed (Participants) | 1089
  Change from BL at Cycle 6 | -1.93 (17.611)
  Change from BL at Cycle 9: number analyzed (Participants) | 1006
  Change from BL at Cycle 9 | 0.87 (17.211)
  Change from BL at Cycle 12: number analyzed (Participants) | 891
  Change from BL at Cycle 12 | 3.03 (17.426)
  Change from BL at Cycle 15: number analyzed (Participants) | 794
  Change from BL at Cycle 15 | 3.33 (18.764)
  Change from BL at Cycle 18: number analyzed (Participants) | 718
  Change from BL at Cycle 18 | 3.80 (18.689)
  Change from BL at Cycle 21: number analyzed (Participants) | 615
  Change from BL at Cycle 21 | 4.06 (18.175)
  Change from BL at Cycle 24: number analyzed (Participants) | 570
  Change from BL at Cycle 24 | 3.59 (19.570)
  Change from BL at Cycle 27: number analyzed (Participants) | 512
  Change from BL at Cycle 27 | 3.14 (20.311)
  Change from BL at Cycle 30: number analyzed (Participants) | 515
  Change from BL at Cycle 30 | 3.75 (18.877)
  Change from BL at Cycle 33: number analyzed (Participants) | 468
  Change from BL at Cycle 33 | 3.58 (20.586)
  Change from BL at Cycle 36: number analyzed (Participants) | 427
  Change from BL at Cycle 36 | 3.16 (18.838)
  Change from BL at Cycle 39: number analyzed (Participants) | 419
  Change from BL at Cycle 39 | 1.66 (19.791)
  Change from BL at Cycle 42: number analyzed (Participants) | 385
  Change from BL at Cycle 42 | 2.08 (20.658)
  Change from BL at Cycle 45: number analyzed (Participants) | 361
  Change from BL at Cycle 45 | 2.22 (20.811)
  Change from BL at Cycle 48: number analyzed (Participants) | 340
  Change from BL at Cycle 48 | 1.51 (21.268)
  Change from BL at Cycle 51: number analyzed (Participants) | 308
  Change from BL at Cycle 51 | 1.95 (20.221)
  Change from BL at Cycle 54: number analyzed (Participants) | 282
  Change from BL at Cycle 54 | 0.52 (20.784)
  Change from BL at Cycle 57: number analyzed (Participants) | 286
  Change from BL at Cycle 57 | 0.54 (20.014)
  Change from BL at Cycle 60: number analyzed (Participants) | 262
  Change from BL at Cycle 60 | 0.20 (21.207)
  Change from BL at Cycle 63: number analyzed (Participants) | 268
  Change from BL at Cycle 63 | 0.61 (21.475)
  Change from BL at Cycle 66: number analyzed (Participants) | 241
  Change from BL at Cycle 66 | 0.44 (20.633)
  Change from BL at Cycle 69: number analyzed (Participants) | 236
  Change from BL at Cycle 69 | -0.75 (21.419)
  Change from BL at Cycle 72: number analyzed (Participants) | 219
  Change from BL at Cycle 72 | -1.16 (21.951)
  Change from BL at Cycle 75: number analyzed (Participants) | 213
  Change from BL at Cycle 75 | -1.14 (21.132)
  Change from BL at Cycle 78: number analyzed (Participants) | 207
  Change from BL at Cycle 78 | 0.11 (20.807)
  Change from BL at Cycle 81: number analyzed (Participants) | 192
  Change from BL at Cycle 81 | -1.03 (20.526)
  Change from BL at Cycle 84: number analyzed (Participants) | 181
  Change from BL at Cycle 84 | -1.67 (21.030)
  Change from BL at Cycle 87: number analyzed (Participants) | 174
  Change from BL at Cycle 87 | 0.62 (21.183)
  Change from BL at Cycle 90: number analyzed (Participants) | 147
  Change from BL at Cycle 90 | 0.00 (22.289)
  Change from BL at Cycle 93: number analyzed (Participants) | 129
  Change from BL at Cycle 93 | 0.99 (21.474)
  Change from BL at Cycle 96: number analyzed (Participants) | 106
  Change from BL at Cycle 96 | 2.36 (21.636)
  Change from BL at Cycle 99: number analyzed (Participants) | 85
  Change from BL at Cycle 99 | 1.36 (23.195)
  Change from BL at Cycle 102: number analyzed (Participants) | 69
  Change from BL at Cycle 102 | 1.20 (21.262)
  Change from BL at Cycle 105: number analyzed (Participants) | 55
  Change from BL at Cycle 105 | 3.13 (20.385)
  Change from BL at Cycle 108: number analyzed (Participants) | 44
  Change from BL at Cycle 108 | 2.22 (23.617)
  Change from BL at Cycle 111: number analyzed (Participants) | 36
  Change from BL at Cycle 111 | -0.48 (22.585)
  Change from BL at Cycle 114: number analyzed (Participants) | 19
  Change from BL at Cycle 114 | -4.42 (22.323)
  Change from BL at Cycle 117: number analyzed (Participants) | 11
  Change from BL at Cycle 117 | -4.96 (16.232)
  Change from BL at Cycle 120: number analyzed (Participants) | 4
  Change from BL at Cycle 120 | -8.64 (13.187)
  Change from BL at Cycle 123: number analyzed (Participants) | 2
  Change from BL at Cycle 123 | -20.94 (2.357)
  Change from BL at End of Treatment: number analyzed (Participants) | 454
  Change from BL at End of Treatment | -1.06 (19.923)
  Change from BL at Day 28 of Follow-Up: number analyzed (Participants) | 568
  Change from BL at Day 28 of Follow-Up | -1.96 (21.201)

54. Secondary Outcome: Change From Baseline in FACT-B Questionnaire Physical Well-Being Subscale Score Over the Course of the Study
Description: The FACT-B questionnaire (version 4) was administered only to female participants to assess quality of life in five subscales: physical, social, emotional, and functional well-being, and breast cancer. For the physical well-being subscale, participants were given a series of 7 statements and were asked to rate how true each statement was for them during the past 7 days on a 5-point scale ranging from 0 (not at all) to 4 (very much). The calculated FACT-B physical well-being subscale score, ranging from 0 to 28, was the sum of the scores for each statement only if at least 50% of items had been answered; the higher the score, the better the quality of life. Baseline was defined as the last non-missing measurement taken prior to first dose of study treatment (including unscheduled assessments). Post-baseline values were summarized for planned visits only.
Time Frame: as for outcome 53
Population: ITT Population: only enrolled female participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1429
Score on a scale
  Baseline (BL): Absolute Value at Visit: number analyzed (Participants) | 1331
  Baseline (BL): Absolute Value at Visit | 20.98 (6.044)
  Change from BL at Cycle 3: number analyzed (Participants) | 1193
  Change from BL at Cycle 3 | -1.13 (5.557)
  Change from BL at Cycle 6: number analyzed (Participants) | 1127
  Change from BL at Cycle 6 | -1.61 (5.994)
  Change from BL at Cycle 9: number analyzed (Participants) | 1033
  Change from BL at Cycle 9 | -0.31 (5.604)
  Change from BL at Cycle 12: number analyzed (Participants) | 919
  Change from BL at Cycle 12 | 0.51 (5.599)
  Change from BL at Cycle 15: number analyzed (Participants) | 816
  Change from BL at Cycle 15 | 0.51 (5.652)
  Change from BL at Cycle 18: number analyzed (Participants) | 734
  Change from BL at Cycle 18 | 0.69 (5.543)
  Change from BL at Cycle 21: number analyzed (Participants) | 631
  Change from BL at Cycle 21 | 0.73 (5.616)
  Change from BL at Cycle 24: number analyzed (Participants) | 581
  Change from BL at Cycle 24 | 0.61 (5.690)
  Change from BL at Cycle 27: number analyzed (Participants) | 526
  Change from BL at Cycle 27 | 0.47 (5.761)
  Change from BL at Cycle 30: number analyzed (Participants) | 523
  Change from BL at Cycle 30 | 0.71 (5.584)
  Change from BL at Cycle 33: number analyzed (Participants) | 483
  Change from BL at Cycle 33 | 0.56 (5.894)
  Change from BL at Cycle 36: number analyzed (Participants) | 437
  Change from BL at Cycle 36 | 0.39 (5.512)
  Change from BL at Cycle 39: number analyzed (Participants) | 429
  Change from BL at Cycle 39 | -0.04 (5.647)
  Change from BL at Cycle 42: number analyzed (Participants) | 396
  Change from BL at Cycle 42 | 0.22 (5.604)
  Change from BL at Cycle 45: number analyzed (Participants) | 370
  Change from BL at Cycle 45 | 0.09 (5.698)
  Change from BL at Cycle 48: number analyzed (Participants) | 346
  Change from BL at Cycle 48 | 0.11 (5.564)
  Change from BL at Cycle 51: number analyzed (Participants) | 319
  Change from BL at Cycle 51 | 0.22 (5.280)
  Change from BL at Cycle 54: number analyzed (Participants) | 292
  Change from BL at Cycle 54 | -0.26 (5.765)
  Change from BL at Cycle 57: number analyzed (Participants) | 296
  Change from BL at Cycle 57 | -0.35 (5.695)
  Change from BL at Cycle 60: number analyzed (Participants) | 269
  Change from BL at Cycle 60 | -0.10 (5.630)
  Change from BL at Cycle 63: number analyzed (Participants) | 275
  Change from BL at Cycle 63 | -0.20 (5.696)
  Change from BL at Cycle 66: number analyzed (Participants) | 246
  Change from BL at Cycle 66 | 0.29 (5.338)
  Change from BL at Cycle 69: number analyzed (Participants) | 243
  Change from BL at Cycle 69 | -0.60 (5.579)
  Change from BL at Cycle 72: number analyzed (Participants) | 224
  Change from BL at Cycle 72 | -0.35 (5.494)
  Change from BL at Cycle 75: number analyzed (Participants) | 218
  Change from BL at Cycle 75 | -0.72 (5.507)
  Change from BL at Cycle 78: number analyzed (Participants) | 213
  Change from BL at Cycle 78 | -0.44 (5.379)
  Change from BL at Cycle 81: number analyzed (Participants) | 197
  Change from BL at Cycle 81 | -0.65 (5.029)
  Change from BL at Cycle 84: number analyzed (Participants) | 186
  Change from BL at Cycle 84 | -0.81 (5.249)
  Change from BL at Cycle 87: number analyzed (Participants) | 181
  Change from BL at Cycle 87 | -0.36 (5.391)
  Change from BL at Cycle 90: number analyzed (Participants) | 153
  Change from BL at Cycle 90 | -0.66 (5.332)
  Change from BL at Cycle 93: number analyzed (Participants) | 134
  Change from BL at Cycle 93 | -0.42 (5.788)
  Change from BL at Cycle 96: number analyzed (Participants) | 110
  Change from BL at Cycle 96 | -0.28 (5.178)
  Change from BL at Cycle 99: number analyzed (Participants) | 88
  Change from BL at Cycle 99 | -0.21 (5.474)
  Change from BL at Cycle 102: number analyzed (Participants) | 72
  Change from BL at Cycle 102 | -0.80 (5.269)
  Change from BL at Cycle 105: number analyzed (Participants) | 57
  Change from BL at Cycle 105 | -0.07 (5.133)
  Change from BL at Cycle 108: number analyzed (Participants) | 45
  Change from BL at Cycle 108 | 0.07 (5.775)
  Change from BL at Cycle 111: number analyzed (Participants) | 37
  Change from BL at Cycle 111 | 0.38 (5.309)
  Change from BL at Cycle 114: number analyzed (Participants) | 20
  Change from BL at Cycle 114 | -1.70 (4.950)
  Change from BL at Cycle 117: number analyzed (Participants) | 12
  Change from BL at Cycle 117 | -1.83 (3.474)
  Change from BL at Cycle 120: number analyzed (Participants) | 4
  Change from BL at Cycle 120 | -2.38 (3.092)
  Change from BL at Cycle 123: number analyzed (Participants) | 2
  Change from BL at Cycle 123 | -5.58 (2.946)
  Change from BL at End of Treatment: number analyzed (Participants) | 465
  Change from BL at End of Treatment | -0.73 (6.366)
  Change from BL at Day 28 of Follow-Up: number analyzed (Participants) | 583
  Change from BL at Day 28 of Follow-Up | -0.95 (6.393)

55. Secondary Outcome: Change From Baseline in FACT-B Questionnaire Social Well-Being Subscale Score Over the Course of the Study
Description: The FACT-B questionnaire (version 4) was administered only to female participants to assess quality of life in five subscales: physical, social, emotional, and functional well-being, and breast cancer. For the social well-being subscale, participants were given a series of 7 statements and were asked to rate how true each statement was for them during the past 7 days on a 5-point scale ranging from 0 (not at all) to 4 (very much). The calculated FACT-B social well-being subscale score, ranging from 0 to 28, was the sum of the scores for each statement only if at least 50% of items had been answered; the higher the score, the better the quality of life. Baseline was defined as the last non-missing measurement taken prior to first dose of study treatment (including unscheduled assessments). Post-baseline values were summarized for planned visits only.
Time Frame: as for outcome 53
Population: ITT Population: only enrolled female participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1429
Score on a scale
  Baseline (BL): Absolute Value at Visit: number analyzed (Participants) | 1329
  Baseline (BL): Absolute Value at Visit | 22.24 (4.993)
  Change from BL at Cycle 3: number analyzed (Participants) | 1189
  Change from BL at Cycle 3 | -0.41 (4.145)
  Change from BL at Cycle 6: number analyzed (Participants) | 1118
  Change from BL at Cycle 6 | -1.09 (4.320)
  Change from BL at Cycle 9: number analyzed (Participants) | 1032
  Change from BL at Cycle 9 | -1.02 (4.728)
  Change from BL at Cycle 12: number analyzed (Participants) | 921
  Change from BL at Cycle 12 | -1.19 (4.846)
  Change from BL at Cycle 15: number analyzed (Participants) | 812
  Change from BL at Cycle 15 | -1.28 (4.949)
  Change from BL at Cycle 18: number analyzed (Participants) | 733
  Change from BL at Cycle 18 | -1.19 (4.986)
  Change from BL at Cycle 21: number analyzed (Participants) | 630
  Change from BL at Cycle 21 | -1.24 (4.881)
  Change from BL at Cycle 24: number analyzed (Participants) | 580
  Change from BL at Cycle 24 | -1.26 (4.856)
  Change from BL at Cycle 27: number analyzed (Participants) | 525
  Change from BL at Cycle 27 | -1.48 (4.994)
  Change from BL at Cycle 30: number analyzed (Participants) | 523
  Change from BL at Cycle 30 | -1.18 (5.107)
  Change from BL at Cycle 33: number analyzed (Participants) | 482
  Change from BL at Cycle 33 | -1.45 (4.852)
  Change from BL at Cycle 36: number analyzed (Participants) | 437
  Change from BL at Cycle 36 | -1.54 (4.953)
  Change from BL at Cycle 39: number analyzed (Participants) | 430
  Change from BL at Cycle 39 | -1.77 (5.066)
  Change from BL at Cycle 42: number analyzed (Participants) | 394
  Change from BL at Cycle 42 | -1.73 (5.154)
  Change from BL at Cycle 45: number analyzed (Participants) | 370
  Change from BL at Cycle 45 | -1.50 (5.238)
  Change from BL at Cycle 48: number analyzed (Participants) | 345
  Change from BL at Cycle 48 | -1.84 (5.475)
  Change from BL at Cycle 51: number analyzed (Participants) | 318
  Change from BL at Cycle 51 | -2.01 (5.657)
  Change from BL at Cycle 54: number analyzed (Participants) | 293
  Change from BL at Cycle 54 | -1.77 (5.236)
  Change from BL at Cycle 57: number analyzed (Participants) | 297
  Change from BL at Cycle 57 | -1.88 (5.117)
  Change from BL at Cycle 60: number analyzed (Participants) | 270
  Change from BL at Cycle 60 | -2.01 (5.528)
  Change from BL at Cycle 63: number analyzed (Participants) | 277
  Change from BL at Cycle 63 | -2.18 (5.278)
  Change from BL at Cycle 66: number analyzed (Participants) | 246
  Change from BL at Cycle 66 | -2.19 (5.586)
  Change from BL at Cycle 69: number analyzed (Participants) | 243
  Change from BL at Cycle 69 | -2.24 (5.434)
  Change from BL at Cycle 72: number analyzed (Participants) | 224
  Change from BL at Cycle 72 | -2.49 (5.846)
  Change from BL at Cycle 75: number analyzed (Participants) | 219
  Change from BL at Cycle 75 | -2.40 (5.777)
  Change from BL at Cycle 78: number analyzed (Participants) | 213
  Change from BL at Cycle 78 | -2.33 (5.676)
  Change from BL at Cycle 81: number analyzed (Participants) | 197
  Change from BL at Cycle 81 | -2.53 (5.609)
  Change from BL at Cycle 84: number analyzed (Participants) | 187
  Change from BL at Cycle 84 | -2.96 (5.624)
  Change from BL at Cycle 87: number analyzed (Participants) | 181
  Change from BL at Cycle 87 | -2.29 (5.487)
  Change from BL at Cycle 90: number analyzed (Participants) | 152
  Change from BL at Cycle 90 | -2.38 (5.355)
  Change from BL at Cycle 93: number analyzed (Participants) | 134
  Change from BL at Cycle 93 | -1.97 (5.102)
  Change from BL at Cycle 96: number analyzed (Participants) | 110
  Change from BL at Cycle 96 | -1.94 (4.831)
  Change from BL at Cycle 99: number analyzed (Participants) | 89
  Change from BL at Cycle 99 | -2.07 (5.316)
  Change from BL at Cycle 102: number analyzed (Participants) | 73
  Change from BL at Cycle 102 | -1.70 (4.258)
  Change from BL at Cycle 105: number analyzed (Participants) | 58
  Change from BL at Cycle 105 | -1.76 (4.074)
  Change from BL at Cycle 108: number analyzed (Participants) | 46
  Change from BL at Cycle 108 | -1.75 (3.387)
  Change from BL at Cycle 111: number analyzed (Participants) | 38
  Change from BL at Cycle 111 | -1.94 (3.663)
  Change from BL at Cycle 114: number analyzed (Participants) | 20
  Change from BL at Cycle 114 | -2.31 (3.386)
  Change from BL at Cycle 117: number analyzed (Participants) | 12
  Change from BL at Cycle 117 | -1.83 (3.600)
  Change from BL at Cycle 120: number analyzed (Participants) | 4
  Change from BL at Cycle 120 | -2.85 (5.485)
  Change from BL at Cycle 123: number analyzed (Participants) | 2
  Change from BL at Cycle 123 | -1.92 (2.946)
  Change from BL at End of Treatment: number analyzed (Participants) | 461
  Change from BL at End of Treatment | -1.29 (4.911)
  Change from BL at Day 28 of Follow-Up: number analyzed (Participants) | 581
  Change from BL at Day 28 of Follow-Up | -1.61 (5.080)

56. Secondary Outcome: Change From Baseline in FACT-B Questionnaire Emotional Well-Being Subscale Score Over the Course of the Study
Description: The FACT-B questionnaire (version 4) was administered only to female participants to assess quality of life in five subscales: physical, social, emotional, and functional well-being, and breast cancer. For the emotional well-being subscale, participants were given a series of 6 statements and were asked to rate how true each statement was for them during the past 7 days on a 5-point scale ranging from 0 (not at all) to 4 (very much). The calculated FACT-B emotional well-being subscale score, ranging from 0 to 24, was the sum of the scores for each statement only if at least 50% of items had been answered; the higher the score, the better the quality of life. Baseline was defined as the last non-missing measurement taken prior to first dose of study treatment (including unscheduled assessments). Post-baseline values were summarized for planned visits only.
Time Frame: as for outcome 53
Population: ITT Population: only enrolled female participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1429
Score on a scale
  Baseline (BL): Absolute Value at Visit: number analyzed (Participants) | 1333
  Baseline (BL): Absolute Value at Visit | 15.08 (4.990)
  Change from BL at Cycle 3: number analyzed (Participants) | 1194
  Change from BL at Cycle 3 | 1.69 (4.219)
  Change from BL at Cycle 6: number analyzed (Participants) | 1124
  Change from BL at Cycle 6 | 1.53 (4.526)
  Change from BL at Cycle 9: number analyzed (Participants) | 1032
  Change from BL at Cycle 9 | 1.64 (4.624)
  Change from BL at Cycle 12: number analyzed (Participants) | 916
  Change from BL at Cycle 12 | 2.02 (4.686)
  Change from BL at Cycle 15: number analyzed (Participants) | 811
  Change from BL at Cycle 15 | 1.98 (4.778)
  Change from BL at Cycle 18: number analyzed (Participants) | 731
  Change from BL at Cycle 18 | 2.03 (4.861)
  Change from BL at Cycle 21: number analyzed (Participants) | 628
  Change from BL at Cycle 21 | 2.17 (4.877)
  Change from BL at Cycle 24: number analyzed (Participants) | 581
  Change from BL at Cycle 24 | 2.19 (5.040)
  Change from BL at Cycle 27: number analyzed (Participants) | 523
  Change from BL at Cycle 27 | 2.21 (5.171)
  Change from BL at Cycle 30: number analyzed (Participants) | 523
  Change from BL at Cycle 30 | 2.17 (4.763)
  Change from BL at Cycle 33: number analyzed (Participants) | 478
  Change from BL at Cycle 33 | 2.21 (5.275)
  Change from BL at Cycle 36: number analyzed (Participants) | 435
  Change from BL at Cycle 36 | 2.32 (5.130)
  Change from BL at Cycle 39: number analyzed (Participants) | 430
  Change from BL at Cycle 39 | 1.99 (5.115)
  Change from BL at Cycle 42: number analyzed (Participants) | 394
  Change from BL at Cycle 42 | 1.96 (5.451)
  Change from BL at Cycle 45: number analyzed (Participants) | 367
  Change from BL at Cycle 45 | 2.25 (5.367)
  Change from BL at Cycle 48: number analyzed (Participants) | 343
  Change from BL at Cycle 48 | 1.82 (5.414)
  Change from BL at Cycle 51: number analyzed (Participants) | 317
  Change from BL at Cycle 51 | 2.32 (5.311)
  Change from BL at Cycle 54: number analyzed (Participants) | 288
  Change from BL at Cycle 54 | 1.84 (5.325)
  Change from BL at Cycle 57: number analyzed (Participants) | 293
  Change from BL at Cycle 57 | 1.80 (5.256)
  Change from BL at Cycle 60: number analyzed (Participants) | 268
  Change from BL at Cycle 60 | 1.59 (5.462)
  Change from BL at Cycle 63: number analyzed (Participants) | 274
  Change from BL at Cycle 63 | 1.70 (5.336)
  Change from BL at Cycle 66: number analyzed (Participants) | 246
  Change from BL at Cycle 66 | 1.52 (5.074)
  Change from BL at Cycle 69: number analyzed (Participants) | 243
  Change from BL at Cycle 69 | 1.83 (5.351)
  Change from BL at Cycle 72: number analyzed (Participants) | 223
  Change from BL at Cycle 72 | 1.56 (5.421)
  Change from BL at Cycle 75: number analyzed (Participants) | 217
  Change from BL at Cycle 75 | 1.58 (5.308)
  Change from BL at Cycle 78: number analyzed (Participants) | 210
  Change from BL at Cycle 78 | 1.72 (5.463)
  Change from BL at Cycle 81: number analyzed (Participants) | 196
  Change from BL at Cycle 81 | 2.01 (5.750)
  Change from BL at Cycle 84: number analyzed (Participants) | 185
  Change from BL at Cycle 84 | 2.06 (5.384)
  Change from BL at Cycle 87: number analyzed (Participants) | 180
  Change from BL at Cycle 87 | 1.97 (5.558)
  Change from BL at Cycle 90: number analyzed (Participants) | 151
  Change from BL at Cycle 90 | 2.08 (5.686)
  Change from BL at Cycle 93: number analyzed (Participants) | 134
  Change from BL at Cycle 93 | 2.17 (5.388)
  Change from BL at Cycle 96: number analyzed (Participants) | 109
  Change from BL at Cycle 96 | 2.40 (5.769)
  Change from BL at Cycle 99: number analyzed (Participants) | 88
  Change from BL at Cycle 99 | 2.30 (6.041)
  Change from BL at Cycle 102: number analyzed (Participants) | 71
  Change from BL at Cycle 102 | 2.07 (5.949)
  Change from BL at Cycle 105: number analyzed (Participants) | 58
  Change from BL at Cycle 105 | 2.58 (5.902)
  Change from BL at Cycle 108: number analyzed (Participants) | 46
  Change from BL at Cycle 108 | 2.34 (6.721)
  Change from BL at Cycle 111: number analyzed (Participants) | 38
  Change from BL at Cycle 111 | 1.19 (7.241)
  Change from BL at Cycle 114: number analyzed (Participants) | 20
  Change from BL at Cycle 114 | 1.55 (7.944)
  Change from BL at Cycle 117: number analyzed (Participants) | 12
  Change from BL at Cycle 117 | 1.33 (4.185)
  Change from BL at Cycle 120: number analyzed (Participants) | 4
  Change from BL at Cycle 120 | 0.75 (2.217)
  Change from BL at Cycle 123: number analyzed (Participants) | 2
  Change from BL at Cycle 123 | -0.50 (2.121)
  Change from BL at End of Treatment: number analyzed (Participants) | 465
  Change from BL at End of Treatment | 0.30 (5.001)
  Change from BL at Day 28 of Follow-Up: number analyzed (Participants) | 585
  Change from BL at Day 28 of Follow-Up | 0.37 (5.193)

57. Secondary Outcome: Change From Baseline in FACT-B Questionnaire Functional Well-Being Subscale Score Over the Course of the Study
Description: The FACT-B questionnaire (version 4) was administered only to female participants to assess quality of life in five subscales: physical, social, emotional, and functional well-being, and breast cancer. For the functional well-being subscale, participants were given a series of 7 statements and were asked to rate how true each statement was for them during the past 7 days on a 5-point scale ranging from 0 (not at all) to 4 (very much). The calculated FACT-B functional well-being subscale score, ranging from 0 to 28, was the sum of the scores for each statement only if at least 50% of items had been answered; the higher the score, the better the quality of life. Baseline was defined as the last non-missing measurement taken prior to first dose of study treatment (including unscheduled assessments). Post-baseline values were summarized for planned visits only.
Time Frame: as for outcome 53
Population: ITT Population: only enrolled female participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1429
Score on a scale
  Baseline (BL): Absolute Value at Visit: number analyzed (Participants) | 1335
  Baseline (BL): Absolute Value at Visit | 16.65 (6.096)
  Change from BL at Cycle 3: number analyzed (Participants) | 1192
  Change from BL at Cycle 3 | -0.47 (4.961)
  Change from BL at Cycle 6: number analyzed (Participants) | 1125
  Change from BL at Cycle 6 | -0.79 (5.437)
  Change from BL at Cycle 9: number analyzed (Participants) | 1032
  Change from BL at Cycle 9 | -0.11 (5.572)
  Change from BL at Cycle 12: number analyzed (Participants) | 915
  Change from BL at Cycle 12 | 0.46 (5.577)
  Change from BL at Cycle 15: number analyzed (Participants) | 814
  Change from BL at Cycle 15 | 0.78 (5.758)
  Change from BL at Cycle 18: number analyzed (Participants) | 732
  Change from BL at Cycle 18 | 0.83 (5.797)
  Change from BL at Cycle 21: number analyzed (Participants) | 629
  Change from BL at Cycle 21 | 0.89 (5.804)
  Change from BL at Cycle 24: number analyzed (Participants) | 583
  Change from BL at Cycle 24 | 0.53 (5.903)
  Change from BL at Cycle 27: number analyzed (Participants) | 523
  Change from BL at Cycle 27 | 0.71 (6.064)
  Change from BL at Cycle 30: number analyzed (Participants) | 524
  Change from BL at Cycle 30 | 0.60 (5.961)
  Change from BL at Cycle 33: number analyzed (Participants) | 478
  Change from BL at Cycle 33 | 0.67 (6.209)
  Change from BL at Cycle 36: number analyzed (Participants) | 436
  Change from BL at Cycle 36 | 0.52 (5.687)
  Change from BL at Cycle 39: number analyzed (Participants) | 430
  Change from BL at Cycle 39 | 0.26 (5.927)
  Change from BL at Cycle 42: number analyzed (Participants) | 393
  Change from BL at Cycle 42 | 0.31 (6.038)
  Change from BL at Cycle 45: number analyzed (Participants) | 368
  Change from BL at Cycle 45 | 0.34 (6.049)
  Change from BL at Cycle 48: number analyzed (Participants) | 344
  Change from BL at Cycle 48 | 0.28 (6.227)
  Change from BL at Cycle 51: number analyzed (Participants) | 319
  Change from BL at Cycle 51 | 0.23 (5.931)
  Change from BL at Cycle 54: number analyzed (Participants) | 289
  Change from BL at Cycle 54 | -0.06 (6.090)
  Change from BL at Cycle 57: number analyzed (Participants) | 294
  Change from BL at Cycle 57 | 0.21 (5.925)
  Change from BL at Cycle 60: number analyzed (Participants) | 268
  Change from BL at Cycle 60 | 0.01 (6.100)
  Change from BL at Cycle 63: number analyzed (Participants) | 275
  Change from BL at Cycle 63 | -0.06 (6.178)
  Change from BL at Cycle 66: number analyzed (Participants) | 247
  Change from BL at Cycle 66 | -0.07 (6.264)
  Change from BL at Cycle 69: number analyzed (Participants) | 243
  Change from BL at Cycle 69 | -0.47 (6.476)
  Change from BL at Cycle 72: number analyzed (Participants) | 224
  Change from BL at Cycle 72 | -0.50 (6.378)
  Change from BL at Cycle 75: number analyzed (Participants) | 217
  Change from BL at Cycle 75 | -0.40 (6.391)
  Change from BL at Cycle 78: number analyzed (Participants) | 211
  Change from BL at Cycle 78 | -0.18 (6.197)
  Change from BL at Cycle 81: number analyzed (Participants) | 197
  Change from BL at Cycle 81 | -0.29 (6.046)
  Change from BL at Cycle 84: number analyzed (Participants) | 186
  Change from BL at Cycle 84 | -0.48 (6.022)
  Change from BL at Cycle 87: number analyzed (Participants) | 180
  Change from BL at Cycle 87 | -0.08 (6.250)
  Change from BL at Cycle 90: number analyzed (Participants) | 152
  Change from BL at Cycle 90 | 0.16 (6.587)
  Change from BL at Cycle 93: number analyzed (Participants) | 135
  Change from BL at Cycle 93 | 0.58 (6.161)
  Change from BL at Cycle 96: number analyzed (Participants) | 111
  Change from BL at Cycle 96 | 1.27 (6.663)
  Change from BL at Cycle 99: number analyzed (Participants) | 89
  Change from BL at Cycle 99 | 0.46 (6.651)
  Change from BL at Cycle 102: number analyzed (Participants) | 73
  Change from BL at Cycle 102 | 0.96 (6.327)
  Change from BL at Cycle 105: number analyzed (Participants) | 59
  Change from BL at Cycle 105 | 1.14 (5.922)
  Change from BL at Cycle 108: number analyzed (Participants) | 46
  Change from BL at Cycle 108 | 1.42 (6.902)
  Change from BL at Cycle 111: number analyzed (Participants) | 38
  Change from BL at Cycle 111 | 0.32 (6.507)
  Change from BL at Cycle 114: number analyzed (Participants) | 20
  Change from BL at Cycle 114 | -0.25 (6.439)
  Change from BL at Cycle 117: number analyzed (Participants) | 12
  Change from BL at Cycle 117 | -0.58 (5.316)
  Change from BL at Cycle 120: number analyzed (Participants) | 4
  Change from BL at Cycle 120 | -2.00 (3.916)
  Change from BL at Cycle 123: number analyzed (Participants) | 2
  Change from BL at Cycle 123 | -5.00 (2.828)
  Change from BL at End of Treatment: number analyzed (Participants) | 463
  Change from BL at End of Treatment | -0.50 (6.132)
  Change from BL at Day 28 of Follow-Up: number analyzed (Participants) | 586
  Change from BL at Day 28 of Follow-Up | -0.70 (6.558)

58. Secondary Outcome: Change From Baseline in FACT-B Questionnaire Breast Cancer Subscale Score Over the Course of the Study
Description: The FACT-B questionnaire (version 4) was administered only to female participants to assess quality of life in five subscales: physical, social, emotional, and functional well-being, and breast cancer. For the breast cancer subscale, participants were given a series of 10 statements and were asked to rate how true each statement was for them during the past 7 days on a 5-point scale ranging from 0 (not at all) to 4 (very much). The calculated FACT-B breast cancer subscale score, ranging from 0 to 40, was the sum of the scores for each statement only if at least 50% of items had been answered; the higher the score, the better the quality of life. Baseline was defined as the last non-missing measurement taken prior to first dose of study treatment (including unscheduled assessments). Post-baseline values were summarized for planned visits only.
Time Frame: as for outcome 53
Population: ITT Population: only enrolled female participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pertuzumab + Trastuzumab + Taxane
Number analyzed (Participants) | 1429
Score on a scale
  Baseline (BL): Absolute Value at Visit: number analyzed (Participants) | 1326
  Baseline (BL): Absolute Value at Visit | 24.98 (6.296)
  Change from BL at Cycle 3: number analyzed (Participants) | 1181
  Change from BL at Cycle 3 | 0.48 (5.101)
  Change from BL at Cycle 6: number analyzed (Participants) | 1117
  Change from BL at Cycle 6 | -0.11 (5.759)
  Change from BL at Cycle 9: number analyzed (Participants) | 1027
  Change from BL at Cycle 9 | 0.52 (5.633)
  Change from BL at Cycle 12: number analyzed (Participants) | 910
  Change from BL at Cycle 12 | 0.89 (5.770)
  Change from BL at Cycle 15: number analyzed (Participants) | 808
  Change from BL at Cycle 15 | 1.16 (6.180)
  Change from BL at Cycle 18: number analyzed (Participants) | 729
  Change from BL at Cycle 18 | 1.30 (6.043)
  Change from BL at Cycle 21: number analyzed (Participants) | 625
  Change from BL at Cycle 21 | 1.30 (5.898)
  Change from BL at Cycle 24: number analyzed (Participants) | 580
  Change from BL at Cycle 24 | 1.39 (6.231)
  Change from BL at Cycle 27: number analyzed (Participants) | 520
  Change from BL at Cycle 27 | 1.17 (6.043)
  Change from BL at Cycle 30: number analyzed (Participants) | 521
  Change from BL at Cycle 30 | 1.34 (5.968)
  Change from BL at Cycle 33: number analyzed (Participants) | 477
  Change from BL at Cycle 33 | 1.34 (6.113)
  Change from BL at Cycle 36: number analyzed (Participants) | 435
  Change from BL at Cycle 36 | 1.33 (6.030)
  Change from BL at Cycle 39: number analyzed (Participants) | 427
  Change from BL at Cycle 39 | 1.12 (6.210)
  Change from BL at Cycle 42: number analyzed (Participants) | 393
  Change from BL at Cycle 42 | 1.11 (6.499)
  Change from BL at Cycle 45: number analyzed (Participants) | 366
  Change from BL at Cycle 45 | 1.13 (6.414)
  Change from BL at Cycle 48: number analyzed (Participants) | 343
  Change from BL at Cycle 48 | 1.00 (6.679)
  Change from BL at Cycle 51: number analyzed (Participants) | 316
  Change from BL at Cycle 51 | 0.99 (6.430)
  Change from BL at Cycle 54: number analyzed (Participants) | 291
  Change from BL at Cycle 54 | 0.76 (6.555)
  Change from BL at Cycle 57: number analyzed (Participants) | 294
  Change from BL at Cycle 57 | 0.70 (6.355)
  Change from BL at Cycle 60: number analyzed (Participants) | 267
  Change from BL at Cycle 60 | 0.80 (6.586)
  Change from BL at Cycle 63: number analyzed (Participants) | 274
  Change from BL at Cycle 63 | 1.32 (6.960)
  Change from BL at Cycle 66: number analyzed (Participants) | 246
  Change from BL at Cycle 66 | 0.74 (6.822)
  Change from BL at Cycle 69: number analyzed (Participants) | 241
  Change from BL at Cycle 69 | 0.54 (6.532)
  Change from BL at Cycle 72: number analyzed (Participants) | 223
  Change from BL at Cycle 72 | 0.50 (7.142)
  Change from BL at Cycle 75: number analyzed (Participants) | 216
  Change from BL at Cycle 75 | 0.85 (6.925)
  Change from BL at Cycle 78: number analyzed (Participants) | 210
  Change from BL at Cycle 78 | 1.22 (6.899)
  Change from BL at Cycle 81: number analyzed (Participants) | 196
  Change from BL at Cycle 81 | 0.27 (7.100)
  Change from BL at Cycle 84: number analyzed (Participants) | 184
  Change from BL at Cycle 84 | 0.55 (6.690)
  Change from BL at Cycle 87: number analyzed (Participants) | 178
  Change from BL at Cycle 87 | 1.17 (6.882)
  Change from BL at Cycle 90: number analyzed (Participants) | 150
  Change from BL at Cycle 90 | 0.51 (7.313)
  Change from BL at Cycle 93: number analyzed (Participants) | 132
  Change from BL at Cycle 93 | 0.30 (7.163)
  Change from BL at Cycle 96: number analyzed (Participants) | 110
  Change from BL at Cycle 96 | 0.65 (6.240)
  Change from BL at Cycle 99: number analyzed (Participants) | 87
  Change from BL at Cycle 99 | 1.19 (6.957)
  Change from BL at Cycle 102: number analyzed (Participants) | 72
  Change from BL at Cycle 102 | 0.56 (6.189)
  Change from BL at Cycle 105: number analyzed (Participants) | 58
  Change from BL at Cycle 105 | 0.68 (6.399)
  Change from BL at Cycle 108: number analyzed (Participants) | 45
  Change from BL at Cycle 108 | 0.19 (6.982)
  Change from BL at Cycle 111: number analyzed (Participants) | 36
  Change from BL at Cycle 111 | 0.01 (6.814)
  Change from BL at Cycle 114: number analyzed (Participants) | 19
  Change from BL at Cycle 114 | -1.67 (5.963)
  Change from BL at Cycle 117: number analyzed (Participants) | 11
  Change from BL at Cycle 117 | -1.56 (5.842)
  Change from BL at Cycle 120: number analyzed (Participants) | 4
  Change from BL at Cycle 120 | -2.17 (6.055)
  Change from BL at Cycle 123: number analyzed (Participants) | 2
  Change from BL at Cycle 123 | -7.94 (7.307)
  Change from BL at End of Treatment: number analyzed (Participants) | 459
  Change from BL at End of Treatment | 0.88 (6.574)
  Change from BL at Day 28 of Follow-Up: number analyzed (Participants) | 576
  Change from BL at Day 28 of Follow-Up | 0.66 (6.477)

ADVERSE EVENTS:
Time Frame: From Baseline until 28 days after last dose of study treatment. The median (full range) duration of exposure to any study treatment was 16.2 (0.0-86.4) months.
Arm/Group | Pertuzumab + Trastuzumab + Taxane
All-Cause Mortality (participants affected / at risk) | 658/1436
Serious Adverse Events (participants affected / at risk) | 535/1436
Other Adverse Events (participants affected / at risk) | 1394/1436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab + Trastuzumab + Taxane (N=1436)
Pneumonia (Infections and infestations) | 26 (30)
Cellulitis (Infections and infestations) | 15 (19)
Urinary tract infection (Infections and infestations) | 15 (15)
Neutropenic sepsis (Infections and infestations) | 10 (10)
Sepsis (Infections and infestations) | 10 (11)
Vascular device infection (Infections and infestations) | 9 (9)
Device related infection (Infections and infestations) | 8 (9)
Respiratory tract infection (Infections and infestations) | 7 (7)
Erysipelas (Infections and infestations) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Influenza (Infections and infestations) | 5 (5)
Lower respiratory tract infection (Infections and infestations) | 5 (5)
Gastroenteritis (Infections and infestations) | 4 (4)
Arthritis bacterial (Infections and infestations) | 3 (3)
Herpes zoster (Infections and infestations) | 3 (3)
Pyelonephritis (Infections and infestations) | 3 (4)
Viral infection (Infections and infestations) | 3 (3)
Bacteraemia (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (4)
Extradural abscess (Infections and infestations) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Neutropenic infection (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Clostridium colitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Dysentery (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (2)
Lung abscess (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Pyomyositis (Infections and infestations) | 1 (2)
Salmonellosis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sinusitis fungal (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 71 (75)
Neutropenia (Blood and lymphatic system disorders) | 47 (56)
Anaemia (Blood and lymphatic system disorders) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 36 (43)
Vomiting (Gastrointestinal disorders) | 7 (8)
Colitis (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 18 (21)
Asthenia (General disorders) | 6 (6)
General physical health deterioration (General disorders) | 5 (7)
Death (General disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Chills (General disorders) | 2 (2)
Mucosal inflammation (General disorders) | 2 (2)
Catheter site inflammation (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Device related thrombosis (General disorders) | 1 (1)
Drug intolerance (General disorders) | 1 (1)
Inflammatory pain (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Nodule (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 8 (8)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (8)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1)
Chemical burns of eye (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (2)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb injury (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (2)
Cardiac failure (Cardiac disorders) | 12 (13)
Atrial fibrillation (Cardiac disorders) | 8 (10)
Atrial thrombosis (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1)
Intracardiac mass (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ejection fraction decreased (Investigations) | 18 (19)
Neutrophil count decreased (Investigations) | 11 (18)
White blood cell count decreased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Computerised tomogram abdomen abnormal (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Neuropsychiatric lupus (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Progressive supranuclear palsy (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1)
Transverse sinus thrombosis (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 7 (9)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 20 (20)
Hypersensitivity (Immune system disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Circulatory collapse (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
B-cell type acute leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (8)
Renal failure (Renal and urinary disorders) | 3 (4)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1)
Psychiatric decompensation (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2)
Pemphigus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Breast haematoma (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Device breakage (Product Issues) | 1 (1)
Device loosening (Product Issues) | 1 (1)
Hypogonadism (Endocrine disorders) | 1 (1)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab + Trastuzumab + Taxane (N=1436)
Diarrhoea (Gastrointestinal disorders) | 974 (2753)
Nausea (Gastrointestinal disorders) | 512 (918)
Vomiting (Gastrointestinal disorders) | 340 (531)
Constipation (Gastrointestinal disorders) | 235 (347)
Stomatitis (Gastrointestinal disorders) | 210 (326)
Abdominal pain (Gastrointestinal disorders) | 206 (314)
Abdominal pain upper (Gastrointestinal disorders) | 149 (187)
Dyspepsia (Gastrointestinal disorders) | 141 (170)
Haemorrhoids (Gastrointestinal disorders) | 79 (92)
Fatigue (General disorders) | 457 (829)
Asthenia (General disorders) | 426 (1123)
Mucosal inflammation (General disorders) | 287 (490)
Pyrexia (General disorders) | 258 (387)
Oedema peripheral (General disorders) | 257 (344)
Influenza like illness (General disorders) | 96 (136)
Pain (General disorders) | 81 (114)
Chills (General disorders) | 75 (84)
Chest pain (General disorders) | 74 (86)
Alopecia (Skin and subcutaneous tissue disorders) | 693 (813)
Rash (Skin and subcutaneous tissue disorders) | 365 (596)
Pruritus (Skin and subcutaneous tissue disorders) | 292 (466)
Dry skin (Skin and subcutaneous tissue disorders) | 167 (208)
Nail disorder (Skin and subcutaneous tissue disorders) | 163 (197)
Erythema (Skin and subcutaneous tissue disorders) | 137 (183)
Onycholysis (Skin and subcutaneous tissue disorders) | 118 (179)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 75 (94)
Headache (Nervous system disorders) | 328 (542)
Neuropathy peripheral (Nervous system disorders) | 328 (537)
Paraesthesia (Nervous system disorders) | 221 (366)
Dizziness (Nervous system disorders) | 205 (271)
Dysgeusia (Nervous system disorders) | 141 (193)
Peripheral sensory neuropathy (Nervous system disorders) | 120 (158)
Taste disorder (Nervous system disorders) | 75 (92)
Neurotoxicity (Nervous system disorders) | 72 (118)
Arthralgia (Musculoskeletal and connective tissue disorders) | 328 (550)
Myalgia (Musculoskeletal and connective tissue disorders) | 284 (476)
Back pain (Musculoskeletal and connective tissue disorders) | 220 (289)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 196 (292)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 195 (248)
Bone pain (Musculoskeletal and connective tissue disorders) | 135 (185)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 128 (157)
Cough (Respiratory, thoracic and mediastinal disorders) | 271 (410)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 263 (360)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 195 (260)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 124 (156)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 100 (135)
Nasopharyngitis (Infections and infestations) | 183 (309)
Urinary tract infection (Infections and infestations) | 180 (294)
Upper respiratory tract infection (Infections and infestations) | 164 (269)
Influenza (Infections and infestations) | 110 (155)
Conjunctivitis (Infections and infestations) | 99 (125)
Rhinitis (Infections and infestations) | 93 (117)
Anaemia (Blood and lymphatic system disorders) | 312 (521)
Neutropenia (Blood and lymphatic system disorders) | 222 (439)
Leukopenia (Blood and lymphatic system disorders) | 84 (162)
Hypertension (Vascular disorders) | 152 (217)
Hot flush (Vascular disorders) | 129 (165)
Lymphoedema (Vascular disorders) | 98 (121)
Decreased appetite (Metabolism and nutrition disorders) | 274 (447)
Hypokalaemia (Metabolism and nutrition disorders) | 76 (122)
Insomnia (Psychiatric disorders) | 157 (183)
Depression (Psychiatric disorders) | 78 (94)
Anxiety (Psychiatric disorders) | 75 (87)
Ejection fraction decreased (Investigations) | 157 (215)
Weight decreased (Investigations) | 98 (115)
Lacrimation increased (Eye disorders) | 169 (220)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT01572038/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT01572038/SAP_001.pdf